

Doc code: BIOSTAT.SAP. 02

Pag. 1 of 115

| <b>Titolo del Protocollo</b> : A 12-weeks open label, non-inferiority trial comparing HnB products vs ECs in terms of efficacy and adoption rates, acceptability, tolerability, and tobacco harm reduction in healthy smokers, not motivated to quit. | Versione: 1.0 26 Settembre 2017 |
|---|---|
| <b>Prodotto</b> : Sigaretta elettronica/HnB (Heat-not-Burn) | Sponsor: AOU Policlinico Vittorio<br>Emanuele - University of Catania<br>Centro per la cura e la prevenzione del<br>tabagismo |
| Contatti: Pasquale Caponnetto - AOU Policlinico Vittorio Emanuele University of Catania Email: p.caponnetto@unict.it - Phone number: (+39) 095.3781537 | |

| PREPARED BY | | | |
|-------------|------------------------|------------|------------------|
| Name | Qualification | Date | Sign |
| Maurizio | Statistician | 08/07/2020 | Mounin flent. |
| Ceracchi | | | Jour Jacob |
| REVIEWED BY | • | • | • |
| Name | Qualification | Date | Sign |
| Valentina | Project Manager | 08/07/2020 | () 0 = 1 10. |
| Granelli | | | Obenius posselli |
| APPROVED BY | | | |
| Name | Qualification | Date | Sign |
| | Sponsor Representative | | |



Doc code: BIOSTAT.SAP. 02

Pag. 2 of 115

# **VERSION HISTORY**

| Version | Date | Description of the Change(s) |
|---|---|---|
| Final 1.0 | 03 January 2020 | First Final version of the document |
| Final 1.1 | 04 June 2020 | Section 4: PP population definition added. |
| | | Section 5.2: description of derived datasets added. |
| | | Sections 6.8 and 7.5: VO2MAX analysis for the Step Test added. |
| | | Section 7: specification of the analysis populations added |
| | | Section 7.1: definition of "Continuous Quitter" added |
| | | Section 7.2.1: Russell Standard analysis included |
| | | Section 7.2.2: section modified |
| | | Section 8: specification of the analysis populations added |
| | | Appendix 1: Index of the TFLs fixed |
| | | All the mock tables fixed. |
| Final 2.0 | 08 July 2020 | Section 4: PP V7 population definition added. |
| | | Section 9.7: new section included. |
| 1 | | Appendix 5: DRM Minute included. |

# INDEX

| 1 | INTRODUCTION | 5 |
|-----|-----------------------------------------------------|----|
| 1.1 | References | 5 |
| 1.2 | List of abbreviations and acronyms | 5 |
| 2 | STUDY DESCRIPTION | 7 |
| 2.1 | Introduction | 7 |
| 2.2 | Study Objectives | 7 |
| 2.3 | Study Design | 88 |
| 2.4 | Product Administered | 88 |
| 2.5 | Study Plan | 8 |
| 3 | SAMPLE SIZE | 8 |
| 4 | ANALYSIS POPULATIONS | 9 |
| 5 | GENERAL INFORMATION FOR THE ANALYSES | 9 |
| 5.1 | Premature discontinuation and missing data managing | 10 |
| 5.2 | Derived datasets | 10 |
| 6 | PATIENTS CHARACTERISTICS AT BASELINE | 10 |
| 6.1 | Patients' Disposition | 10 |
| 6.2 | Inclusion and Exclusion criteria | 10 |
| 6.3 | B Demographics and smoking habits | 11 |



Doc code: BIOSTAT.SAP. 02

Pag. 3 of 115

| 6.4 | Medical History11 |
|-------|--------------------------------------------------------------------|
| 6.5 | Patients' Characteristics and Vital Signs at Baseline11 |
| 6.6 | Urine collection and storage11 |
| 6.7 | Fagestorm test for nicotine dependence11 |
| 6.8 | Step test12 |
| 6.9 | Device delivery12 |
| 7 ST | ATISTICAL ANALYSES OF THE EFFICACY ENDPOINTS12 |
| 7.1 | Analysis of primary endpoint12 |
| 7.2 | Analysis of secondary endpoints12 |
| 7.2.1 | Smoking reduction derived from the use of HnB and EC13 |
| 7.2.2 | Adoption rate and adherence to product use13 |
| 7.2.3 | Modified Cigarette Evaluation Questionnaire14 |
| 7.2.4 | Smoking Cue Appeal Questionnaire14 |
| 7.2.5 | Intention To Use Questionnaire (ITUQ)14 |
| 7.2.6 | Risk Perception (PRI-P CC)14 |
| 7.2.7 | Risk Perception (PRI-P RRP)15 |
| 7.2.8 | Device Delivery15 |
| 7.3 | Biomarker of Biological Exposure15 |
| 7.4 | EQ-5D15 |
| 7.5 | Step test by visit |
| 8 ST | ATISTICAL ANALYSES OF SAFETY ENDPOINTS16 |
| 8.1 | Extent of Exposure and study duration16 |
| 8.2 | Adverse Events16 |
| 8.3 | Vital signs17 |
| 8.4 | End study information17 |
| 9 DI | ESCRIPTION OF THE STATISTICAL REPORT AND GENERAL FORMAT OF TFLS 17 |
| 9.1 | Presentation of the Data17 |
| 9.2 | Tables, Graphs and Listings Layout18 |
| 9.3 | General Description of the Statistical Report (SR)19 |



Doc code: BIOSTAT.SAP. 02

Pag. 4 of 115

| 9.4 | Responsibilities | 19 |
|-----|-------------------------------------|----|
| 9.5 | Structure of the Statistical Report | 20 |
| 9.6 | Format of the Statistical Report | 20 |
| 9.7 | Decision taken during the DRM | 20 |
| 10 | APPENDIX | 21 |



Doc code: BIOSTAT.SAP. 02

Pag. 5 of 115

#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the study Protocol Final Version (dated September 26, 2017). The main objective of this document is to provide guidance for the production of the analyses of all the variables included in the Database of the study which will be frozen when the last data is validated in accordance with the Fullcro's SOPs.

This document will also provide guidance for the production of the Statistical Report (SR), the in-text tables, the in-text listings and the Tables/Figures/Listings (TFLs) which will be part of the SR as Appendices (they will regard the data of all patients and all variables included in the Database).

The Statistical analysis will begin once the data validation is complete and will proceed according to this plan. In case of deviations from this SAP, explanations in the Statistical Report (SR) will be provided.

This document refers to the analysis of all the variables included in the Clinical Data Base.

All details on the decisions made during the Data Review Meeting (DRM) will be described in an ad hoc section in Version 2.0 of the present document that will be produced before the Database freezing.

#### 1.1 References

- ✓ ICH E6 R1 Guideline GCP
- ✓ SOP\_DM 04\_Convalida dei sistemi
- ✓ SOP\_DM\_03 Data Management
- ✓ SOP\_IT\_01 Gestione dell'infrastruttura IT

#### 1.2 List of abbreviations and acronyms

AE Adverse Event

BoBE Biomarkers of Biological Effects

BP Blood Pressure

DRM Data Review Meeting

EC Electronic Cigarette

eCO Exhaled breath Carbon monoxide

GCP Good Clinical Practice

HnB Heat-not-Burn

HR Heart Rate

ITUQ Intent to use questionnaire



Doc code: BIOSTAT.SAP. 02

Pag. 6 of 115

LOCF Last Observation Carried Forward

mCEQ Modified Cigarette Evaluation Questionnaire

PT Preferred Term

SR Statistic Report

SAE Serious Adverse Event

SOC System Organ Class



Doc code: BIOSTAT.SAP. 02

Pag. 7 of 115

#### 2 STUDY DESCRIPTION

#### 2.1 Introduction

This is a 12-weeks, open label, non-inferiority trial comparing HnB products vs. ECs in terms of efficacy, adoption rate and acceptability, tolerability, and tobacco harm reduction in healthy smokers, not motivated to quit, randomized (1:1) to switch to one of these products. Evaluation of efficacy, adoption rates, acceptability and tolerability will be also recorded at 24 weeks (follow-up).

#### 2.2 Study Objectives

The primary objective of this study is to compare the efficacy of HnB and EC, in terms of quit rates at week 12, by self-reporting abstinence from classic cigarette [validated by an Exhaled breath Carbon monoxide (eCO) measurement ≤10ppm)].

The secondary objectives are:

- to compare the smoking reduction derived from the use of HnB and EC, intended as a 50% reduction in the number of conventional cigarette/day at week 12, defined through selfreporting;
- 2) to compare the adoption rate, and adherence to product use [by collecting (empty) refill bottles and used heathsticks on a daily basis, verified by a study diary filled daily by the subject];
- 3) to compare the acceptability of HnB and of EC, through the assessment of product satisfaction, risk perception, effects on craving and nicotine withdrawal, product preferences, subjective and sensorial effects by:
  - a) Modified Cigarette Evaluation Questionnaire (mCEQ) adapted for EC and HnB users;
  - b) three of 8 items of "Smoking Cue Appeal" adapted for EC and HnBusers;
  - c) "Intent to use questionnaire" (ITUQ) items 4-6;
  - d) PRI-P CC Perceived Health Risk scale (for classic cigarette)
  - e) PRI-P RRP Perceived Health Risk scale (for reduced risk products)
  - f) percentage of choice of a particular subtype of heatstick (HnB) or e-liquid.
- 4) to compare the tolerability of HnB and EC, in terms of: self-reported adverse and serious adverse events by study participants, vital signs (BP, HR and body weight) measurements.
- 5) to compare the tobacco harm reduction between HnB and EC, in terms of:
  - a) changes in Biomarkers of Biological Effects (BoBE) such as: eCO in the exhaled breath (i.e. eCO), step test values;



Doc code: BIOSTAT.SAP. 02

Pag. 8 of 115

b) measurement of 14 selected Biomarkers of Exposure (BoE) in spot urine samples of study participants:

1 tobacco-specific nitrosamine, total NNAL (NNK); 8 volatile organic toxicants (derivates of mercapturic acid, MA): 2-hydroxyethylmercapturic acid (HEMA) also known as ethylene oxide, 2-hydroxy-3-butenyl- mercapturic acid and isomers (MHBMA) also known as 1,3butadiene, 3-hydroxy-1-methyl propyl- mercapturic acid (HMPMA) also known as crotonaldehyde, 3-hydroxypropylmercapturic acid (3-HPMA) also known as acrolein, Sphenylmercapturic acid (S-PMA) also known as benzene, 2-carbamoylethylmer- capturic acid (acrylamide mercapturic acid (AAMA) also known as acrylamide (AAMA and GAMA), cyanoethylmercapturic acid (CEMA) also known as acrylonitrile, hydroxypropylmercapturic acid (2-HPMA) also known as propylene oxide; 4 polycyclic aromatic hydrocarbons: naphthalene, fluorine, phenanthrene, pyrene (1-OHP); cotinine; creatinine.

- c) self-perception of "Tobacco Harm Reduction process" through changes in quality of life scores (EQ-5Dquestionnaire);
- 6) to compare the reliability of HnB and EC, in terms of incidence and kind of malfunctioning events, through self-reporting.

#### 2.3 Study Design

This is a 12-weeks, open label, non-inferiority trial.

#### 2.4 Product Administered

Participants randomized in study group with HnB (group A) will receive one iQOS kit and a 12 weeks supply of heatsticks; those in study with EC (group B) will receive one JustFog Starter Kit and a 12 weeks supply of e-liquids.

#### 2.5 Study Plan

This study has been structured considering a Screening visit (V0), a Baseline visit (V1), a week 1 visit, a week 2 visit, a week 4 visit, a week 8 visit, a week 12 visit. A prospective evaluation of efficacy, adoption rates, acceptability and tolerability will be also recorded at 24-weeks, through a follow-up visit (V7).

#### 3 SAMPLE SIZE



Doc code: BIOSTAT.SAP. 02

Pag. 9 of 115

Sample size determination (better detailed in the study protocol) for no-inferiority testing is based on the assumptions that:

- 1) expected quit rates based on most recent EC literature is about 20-25% and
- 2) that differences in quit rates between products under investigation should not exceed 10-15% (as per non- inferiority definition).

For sample size definition, Farrington-Manning Score Test for Proportion Difference was used, assuming:

- asymptotic normal distribution, upper one-tailed
- alpha 0.05
- nominal power 0.80

Thus:

- Null Proportion Diff. -0.15
- Ref Proportion 0.25
- N per group: 104

According to these hypotheses the required number of participants per study arm was 104. Hence 220 participants, 110 per group, had to be included.

#### 4 ANALYSIS POPULATIONS

In the study protocol the analysis populations were not defined.

As for the safety analyses

the **Safety population**, defined as all the subject who assumed at least one dose of the product, will be considered for the safety analyses.

As for the efficacy analyses

The **Intention-To-treat** population, defined as all the subjects who assumed at least one dose of the study product and had at least one observation after the baseline, will be considered for all the other analyses.

The Per-Protocol population, defined as all the subjects that completed all the visits.

The **Per-Protocol V7** population (see DRM Minute in Appendix 5), defined as all the subjects that completed all the visits, included the Follow-up visit (Visit 7).

#### 5 GENERAL INFORMATION FOR THE ANALYSES



Doc code: BIOSTAT.SAP. 02

Pag. 10 of 115

According to the study protocol the statistical analysis will be descriptive in nature.

All the data will be described using standard descriptive statistics, i.e. n, missing, mean, standard deviation, (25th, 50th, 75th) percentiles for numerical variables. As for the categorical variables, frequency tables with count and percentage will be used. In the core of the Statistical Report, the continuous variables will be presented as mean values ± standard deviation (SD) or median value and interquartile range [IQR], and categorical variables as numbers and percentages. The descriptive analyses will be presented by group. As indicated in the study protocol, for the primary endpoint, the quit rate at 3 months in the experimental study group will be calculated with a non-inferiority threshold of 15%. The quit rates will be evaluated on an intention-to-treat basis: subjects known to have failed will be considered as treatment failures in the primary analysis along with subjects lost to follow-up.

All the analyses will be performed using SAS® Vers. 9.4.

#### 5.1 Premature discontinuation and missing data managing

Patients with missing values will not be excluded from the analysis, their data will not be replaced; frequency of missing data will be given for all analyzed variables. For possible inferential analyses, the LOCF (Last Observation Carried Forward) will be adopted.

#### 5.2 Derived datasets

At the moment of the preparation of the present SAP, three derived dataset is forecasted to be created, i.e. the one containing the MedDRA codes for the Adverse Events, the one containing the information about the adherence to the device and the one containing the analysis populations, that will be prepared after the database freezing. In case additional derived dataset will be needed during the analysis phase, details will be provided in the Statistical Report.

#### **6 PATIENTS CHARACTERISTICS AT BASELINE**

### 6.1 Patients' Disposition

The patients' enrolment will be summarized (Appendix 2: Table D.1) and listed (Appendix 3: Listing D.1). Enrolled, completed and not completed patients, including the reasons, will be summarized with frequency and percentages.

#### 6.2 Inclusion and Exclusion criteria



Doc code: BIOSTAT.SAP. 02

Pag. 11 of 115

The data of the Inclusion and exclusion criteria for all the screened patients will be listed (Appendix 3: Listings D.2 and D.3).

#### 6.3 Demographics and smoking habits

The following demographic and baseline variables will be analyzed: age, gender at birth and education (Appendix 2: Table D.2a). As for the smoking habits, a dedicated table, in which details are presented as summary and frequency tables, will be prepared. Number of cigarettes per day will be summarized (Appendix 2: Table D.2b).

These data will also be listed (Appendix 3: Listing D.4, Listing D.5).

#### 6.4 Medical History

The medical conditions will be coded with the MedDRA dictionary (last available version) and be analyzed as previous and present Medical History using the variable "Ongoing" for creating the two sets of data. The past and present incidence of the different conditions by system organ class and preferred term will be described with frequencies and percentages (Appendix 2: Tables D.3 and D.4a). Present Medical History is defined "In treatment" if the disease is still being treated at the time of the signing of the informed consent and "Not in treatment" otherwise. Present Medical History In treatment and Not in treatment will be summarized through further tables. (Appendix 2: Tables D.4b and D.4c)

These data will also be listed (Appendix 3: Listings D.6, D.7, D.8, D.9).

#### 6.5 Patients' Characteristics and Vital Signs at Baseline

The values of each vital sign variable, i.e. Height, Weight, BMI, FatM, FatP, Total Body Water, Fat Free Mass, Body Muscle Mass, Body Bone Mass, Metabolica Age, Visceral Fat, PAS, PAD and HR will be summarized at baseline in each group through n, missing, mean, standard deviation, (25th, 50th, 75th) percentiles (Appendix 2: Table D.5). These data will also be listed (Appendix 3: Listing S.2).

#### 6.6 Urine collection and storage

Urine collection and storage will be summarized in each group with frequency table regarding to the device given to the subject and with descriptive statistics for the containers delivered (Appendix 2: Table D.6). These data will also be listed (Appendix 3: Listing D.10).

#### 6.7 Fagestorm test for nicotine dependence



Doc code: BIOSTAT.SAP. 02

Pag. 12 of 115

The results of the Fagestorm test for nicotine dependence (FTCD) will be presented as frequencies and percentages for the single questions and total scores derived from the questionnaire through n, missing, mean, standard deviation and 25th, 50th, 75th percentiles (Appendix 2: Table D.7). These data will also be listed (Appendix 3: Listing D.11).

#### 6.8 Step test

The values of Step Test, i.e Baseline, Step 1 to 5 and will be summarized by HR and SpO2 in each group through n, missing, mean, standard deviation and 25th, 50th, 75th percentiles (Appendix 2: Table D.8a). The other items at baseline, i.e. Baseline condition recovery time, Stop time and V02MAX (see Section 7.5 for the definition) will be summarized similarly (Appendix 2: Table D.8b). These data will also be listed (Appendix 3: Listing D.12)

#### 6.9 Device delivery

The data of the device delivery regarding the preferred flavor of chopstick chosen, the device's functioning and the patient training for the device will be summarized in each group through frequency tables for all screened subjects (Appendix 2: Table D.9) and will be listed (Appendix 3: Listings D.13).

#### 7 STATISTICAL ANALYSES OF THE EFFICACY ENDPOINTS

The analyses od the primary and secondary endpoints will be carried out of both the ITT and PP populations. Moreover, as for the Step Test and the Quality of Life (i.e. EQ-5D), a further analysis in the subpopulation od the "Continuous Quitter" will be presented.

#### 7.1 Analysis of primary endpoint

The primary endpoint aims to compare the efficacy of HnB and EC in terms of quit rates at week 12 by means a non-inferiority threshold of 15%.

A "Continuous Quitter" is defined as a subject who has a number of conventional cigarette/day equal to zero from Visit 4 to Visit 6. The Farrington-Manning Score Test for Proportion Difference will be used for comparing the quit rates of the two groups. The SAS® PROC FREQ with the METHOD=FM option will be used. The quit rates of the two groups, along with the relevant 95% Confidence Intervals, will be summarized in Table E.1 (Appendix 2).

#### 7.2 Analysis of secondary endpoints



Doc code: BIOSTAT.SAP. 02

Pag. 13 of 115

The secondary endpoints refer to the smoking reduction, the compliance to the study product and the acceptability of HnB or EC. The analyses to be performed on the smoking reduction and the adoption rate will be presented in sections 7.2.1 and 7.2.2 respectively. As for the latter, the endpoint will be analyzed through the product satisfaction, the risk perception, the effects on craving and nicotine withdrawal, the product preferences, the subjective and sensorial effects and presented in the sections from 7.2.3 to 7.2.8. In sections 7.3 and 7.4 the results of the analyses on the EQ-5D and the step test by visit will be presented.

#### 7.2.1 Smoking reduction derived from the use of HnB and EC

The smoking reduction derived from the use of HnB and EC, will be computed at each visit. The analysis will be presented considering both the definition of "Reducer" included in the study protocol and the so called "Russell Standard" (clinical) for outcome assessment in clinical trials of smoking cessation treatments.

As for the protocol definition, a subject will be classified as "Reducer" if at least a 50% reduction in the number of conventional cigarette/day at each visit will be observed. The results will be summarized as frequency table. The comparison between the two groups will be performed at each visit with the chi-square test. The results will be included in Table E.2a (Appendix 2).

As for the Russell Standard analysis, due to the fact that the study endpoint was a 12 weeks, a small deviation was adopted. In fact, the timepoint considered in the Russell Standard is 52 week. In our case, the 12 week and the 24 week (i.e. the Follow-up observation) will be considered for the analysis. The results will be included in Table E.2b (Appendix 2).

## 7.2.2 Adoption rate and adherence to product use

The adoption rate and adherence to the product use will be analyzed on the basis of the subject's diary. The Sponsor will collect information relevant to the number of days of abservation (i.e. last visie day – Informed Consent day) and the total of days of the device use. Those information will be collected in a derived dataset. The adherence to the producet will be computed in term of rate according to the following formula:

$$Rate = \frac{Total \; days \; of \; device \; use}{Total \; days \; of \; study \; observation}$$

A subject is defined as "compliant" if the rate is at least a 90%. The comparison between the two groups will be performed with the chi-square test. The results will be included in Table E.3 (Appendix 2).



Doc code: BIOSTAT.SAP. 02

Pag. 14 of 115

#### 7.2.3 Modified Cigarette Evaluation Questionnaire

The modified Cigarette Evaluation Questionnaire (mCEQ) will be presented as descriptive summary table by visit. Acceptability of HnB and of EC will be analized through the assessment of several questionnaires. The analyses will be presented in three multi-item domains (i.e. Smoking Satisfaction, Psychological Reward and Avversion) and two single-item domains (i.e. Cravin Reduction and Enjoiment of Respiratory Tract Sensation). Changes from the Baseline Visit to all the subsequent study visits will be also generated. The results will be included in Table E.4a1 (Appendix 2).

The t-test will be carried out on the differences at final visit to baseline. In case the normality assumption is not verified, the corresponding non parametric test will be adopted. The results will be included in Table E.4a2 (Appendix 2). These data will also be listed (Appendix 3: Listing E.2).

#### 7.2.4 Smoking Cue Appeal Questionnaire

The Smoking Cue Appeal Questionnaire will be presented as frequency table of the scores for each question included in the questionnaire. Each table will compare, for each visit in which the questionnaire was administered, the Hnb group and the EC group frequency of answers (Table E.4b1).

The t-test will be carried out on the differences at final visit to baseline. In case the normality assumption is not verified, the corresponding non parametric test will be adopted (Table E.4b2). These data will also be listed (Appendix 3: Listing E.3).

#### 7.2.5 Intention To Use Questionnaire (ITUQ)

Intention To Use Questionnaire (ITUQ) will be presented as frequency table of the scores for each question included in the questionnaire. Each table will compare, for each visit in which the questionnaire was administered, the Hnb group and the EC group frequency of answers (Table E.4c1).

The t-test will be carried out on the differences at final visit to baseline. In case the normality assumption is not verified, the corresponding non parametric test will be adopted (Table E.4c2). These data will also be listed (Appendix 3: Listing E.4).

#### 7.2.6 Risk Perception (PRI-P CC)

Risk Perception (PRI-P CC) Questionnaire will be presented as frequency table of the scores for each question included in the questionnaire. Each table will compare, for each visit in which the questionnaire was administered, the Hnb group and the EC group frequency of answers (Table E.4d1).



Doc code: BIOSTAT.SAP. 02

Pag. 15 of 115

The t-test will be carried out on the differences at final visit to baseline. In case the normality assumption is not verified, the corresponding non parametric test will be adopted (Table E.4d2). These data will also be listed (Appendix 3: Listing E.5).

#### 7.2.7 Risk Perception (PRI-P RRP)

Risk Perception (PRI-P RRP) Questionnaire will be presented as frequency table of the scores for each question included in the questionnaire. Each table will compare, for each visit in which the questionnaire was administered, the Hnb group and the EC group frequency of answers (Table E.4e1)

The t-test will be carried out on the differences at final visit to baseline. In case the normality assumption is not verified, the corresponding non parametric test will be adopted Table E.4e2). These data will also be listed (Appendix 3: Listing E.6).

#### 7.2.8 Device Delivery

Device delivery will be summarized with frequency table for each group. The results will be included in Table E.4f. These data will also be listed (Appendix 3: Listing D.9).

#### 7.3 Biomarker of Biological Exposure

Exhaled breath Carbon monoxide (eCO) will be summarized by timepoint using descriptive summaries as described in Section 5. The parameter will be measured across all the study visits. Changes from the Baseline Visit to all the subsequent study visits will be also generated. Table E.5 will include the summaries of the data by group. The t-test will be carried out on the changes from baseline to last visit. In case the normality assumption is not verified, the corresponding non parametric test will be adopted.

#### 7.4 EQ-5D

The Euro Quality of Life Questionnaire (EQ-5D) will be presented as descriptive summary table by visit. Acceptability of HnB and of EC will be analized through the assessment of several questionnaires. The analyses will be presented throught the five dimensions (i.e. Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression) and a Visual Analogue Scale (EQ VAS). Changes from the Baseline Visit to all the subsequent study visits will be also generated. The results will be included in Table E.6 (Appendix 2).

The t-test will be carried out on the differences at final visit to baseline. In case the normality assumption is not verified, the corresponding non parametric test will be adopted. The results will be



Doc code: BIOSTAT.SAP. 02

Pag. 16 of 115

included in Table E.4a2 (Appendix 2). These data will also be listed (Appendix 3: Listing E.1). The analysis will be presented by all subjects and "Continuous Quitters".

#### 7.5 Step test by visit

The Step test data will be presented as descriptive summary table by visit. The seven items regarding Heart Rate and Oxygen Saturation (i.e. Baseline, Step 1 to 5 and Baseline condition recovery time) will be analysed by HR and SpO2. The two items, (i.e. Stop time and V02MAX, will by analysed using the same methods (Table E.7a). In details, the latter, is the result of the so called "Chester Step Test" who was computed for each subject at site and reported in the eCRF.

An inferential analysis will be carried out on the changes from baseline by item. The results will be presented in Table E.7b. The data will also be listed (Appendix 3: Listing D.8). The analysis will be presented by all subjects and "Continuous Quitters".

#### 8 STATISTICAL ANALYSES OF SAFETY ENDPOINTS

The Safety will be evaluated on all the subjects in the study through the analysis of the Adverse Events (AEs), i.e. those events, occurred during the study, which could be related or not related with the devices, and the Vital Signs.

No methods for replacing missing values will be applied. The Safety population will be considered for this analysis, therefore all the listings will be built with reference to the full set of enrolled patients. As for the Vital Signs, a further analysis in the subpopulation od the "Continuous Quitter" will be presented.

#### 8.1 Extent of Exposure and study duration

The study duration (from Baseline to last Visit) will be summarized in Table S.1 and listed in term of baseline date, final visit date and time interval in days in Listing S.1.

#### 8.2 Adverse Events

Adverse Events will be coded using the MedDRA dictionary (last version available). All the events (i.e., all the conditions which started or deteriorated after the Informed Consent signing) observed during the study will be listed (Listing S.2).

The following summary tables (N, %), replied by Group, will be presented:

✓ Overview of AEs: number of subjects with any AEs, study product related AEs, serious AEs, study product related serious AEs, AEs leading to withdrawal, AEs leading to death (Table S.2a).



Doc code: BIOSTAT.SAP. 02

Pag. 17 of 115

- ✓ Incidence of AEs by SOC and PT (Table S.2b).
- ✓ Incidence of serious AEs by SOC and PT (Table S.2c)
- ✓ Incidence of study treatment related AEs (defined as suspected with respect to product relationship in the opinion of the Investigator) by SOC and PT (Table S.2d).
- ✓ Incidence of AEs leading to study withdrawal by SOC and PT (Tables S.2e).
- ✓ Incidence of AEs by severity and by SOC and PT (Table S.2f).

#### 8.3 Vital signs

Each Vital Sign, i.e. Weight, Height (at baseline only), BMI, Body Fat (FatM and FatP) Total Body Water, Fat Free Mass, Bone Body Mass, Matabolic Age, Visceral Fat, PAS, PAD and HR will be summarized by timepoint using descriptive summaries as described in Section 5.

All the variables will be measured across all the study visits. Changes from the Baseline Visit to all the subsequent study visits will be also generated.

Table S.3 will include the summaries of the Vital Signs by group. A listing will be also produced (Listing S.2).

#### 8.4 End study information

Table S.4 (Appendix 2) will include all the information recorded in the End Study Form of the eCRF, i.e. completeness of the study and frequency table of the reasons for the study interruption. As for the study duration (variable "End Study Date") the analysis will be presented in Table S.1 (see Section 9.1). The data will also be listed in Listing S.3 (Appendix 3).

#### 9 DESCRIPTION OF THE STATISTICAL REPORT AND GENERAL FORMAT OF TFLS

#### 9.1 Presentation of the Data

Tables and listings will be produced in accordance with the principles outlined by the ICH E3 guideline "Note for Guidance on Structure and Content of Clinical Study Report" (CPMP/ICH/137/95).

Quantitative variables will be summarized using the SAS UNIVARIATE or SUMMARY procedures.

Categorical variables will be summarized using the SAS FREQ procedure.

Tables and listings will be produced in accordance with the principles outlined by the ICH E3 guideline and numbered as follows (where n is a sequential number):



Doc code: BIOSTAT.SAP. 02

Pag. 18 of 115

- ✓ Table D.n/Listing Dn for the Baseline characteristics and data collected during the visits other than the Safety ones;
- ✓ Table E.n for the Efficacy data (the Efficacy data will be listed in one of the other three set
  of listings);
- ✓ Table S.n/Listing S.n for the Safety data.

#### 9.2 Tables, Graphs and Listings Layout

The statistical analyses will be performed by the Biostatistician in charge in Fullcro S.r.l.. All tables, figures and listings of the Statistical Report will be generated using the software package SAS® Ver. 9.4.

As for the format of the SAS® outputs (tables and listings), all the pages will contain the following information:

- ✓ Protocol identification.
- ✓ Name of the Sponsor.
- ✓ Specification of document version.
- ✓ Date when the output was generated.

In addition, the following recommendations shall be fulfilled:

- ✓ titles should be fully explicative for the content of the tables/listings;
- ✓ all abbreviations used in any part of the output must be defined in footnotes.

As for character and spacing of the SAS® outputs, the following recommendations shall be fulfilled:

- ✓ SAS Monospace, Size: 8 or 7 (7 or 6 for listings);
- ✓ Margins (for both vertical and horizontal outputs):

Upper 2.5 cm;

Lower 1.0 cm;

Left 2.5 cm;

Right 1.0 cm.

Post-text tables and post-text listings will be included as appendices in the SR.

The post-text tables will be numbered according to presented in the list included in Appendix 1.

The rule for numbering the post-text listings will be as for post-text tables, but a prefix PL will be added.



Doc code: BIOSTAT.SAP. 02

Pag. 19 of 115

#### 9.3 General Description of the Statistical Report (SR)

The Statistical Report (SR) of this study will follow the recommendations given in the guideline ICH topic E3.

American English will be used for writing the SR.

The core of the SR will be written with Microsoft Word<sup>®</sup>; all data summaries (tables) and listings will be prepared by using SAS<sup>®</sup> Version 9.4. In-text tables will be generated with Word. A complete list of the in-text tables is not provided in this document. However, the standard format of these tables must be compliant with the sample illustrated below.

Panel 1: Sample of in-text tables

Table # Sample of in-text tables

| Variable | Group HnC | Group EC |
|---|---|---|
| Continuous variable (unit): | | |
| N | XX | XX |
| Missing | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Q1 – Q3 | xx.x - xx.x | xx.x - xx.x |
| Categorical variable – n (%): | Categorical variable – n (%): | |
| Class 1 | xx (xx.x) | xx (xx.x) |
| Class 2 | xx (xx.x) | xx (xx.x) |
| Class k | xx (xx.x) | xx (xx.x) |

Source: Post-text table # and/or listing #

It is mandatory that every in-text table be cross-referenced with the corresponding post-text tables and listings. In addition, the titles must be auto-explicative and all acronyms must be described in footnotes. When relevant, the time of assessment must be specified.

#### 9.4 Responsibilities

The SR of the present study will be written by the Biostatistician in charge in Fullcro S.r.l. and approved by the Sponsor's representative.



Doc code: BIOSTAT.SAP. 02

Pag. 20 of 115

#### 9.5 Structure of the Statistical Report

The SR will be divided in sections, titled and numbered.

#### 9.6 Format of the Statistical Report

All the pages of the SR core (text) should contain the following information:

- ✓ Protocol identification;
- ✓ Page number;
- ✓ Name of the Sponsor;
- ✓ Specification of document version and date;
- ✓ Information on the level of restriction.

As for character and spacing of the SR core (text), the following recommendations shall be fulfilled:

- ✓ Century Gotic (type size 10);
- ✓ Line spacing 1.5;
- ✓ Justified;
- ✓ Margins as for vertical format:
  - Upper 4.0 cm;
  - Lower 4.2 cm;
  - Left 2.5 cm;
  - Right 2.0 cm.
- ✓ Margins as for horizontal format:
- ✓ Upper 3.5 cm;
- ✓ Lower 2.0 cm;
- ✓ Left 4.2 cm;
- ✓ Right 4.0 cm.
- √ Header 2.0 cm (from upper edge of page);
- ✓ Footer 2.5 cm (from lower edge of page).

#### 9.7 Decision taken during the DRM

As described in the Minute included in Appendix 5, on the 10<sup>th</sup> June 2020 the Data Review Meeting of the study was held in call conference manner. All the decision taken were reported in the Minute. The main decision regarded the analysis population definition. All the protocol violations were evaluated, therefore the following populations were approved by the team:

Population **Safety**: 220



Doc code: BIOSTAT.SAP. 02

Pag. 21 of 115

Population Intention-To-Treat: 217

Population **Per-Protocol**: 193

Population **Per-Protocol V7**: 177

## 10 APPENDIX

Appendix 1 List of TLFs

Appendix 2 Mock Tables: Tables
Appendix 3 Mock Table: Listings
Appendix 4 Study Flow Chart
Appendix 5 DRM Minute



Doc code: BIOSTAT.SAP. 02

Pag. 22 of 115

# APPENDIX 1 List of Tables/Listings to be generated for the Statistical Report



Doc code: BIOSTAT.SAP. 02

Pag. 23 of 115

| Table number | Baseline Characteristics - Table title |
|---|---|
| Table D.1 | Patients Accountability by group |
| Table D.2a | Summary of Demographic and Screening/Baseline Characteristics by group |
| Table D.2b | Summary of Smoking Information at Screening/Baseline by group |
| Table D.3 | Summary of Past Medical History by group |
| Table D.4a | Summary of Present Medical History by group |
| Table D.4b | Summary of Present Medical History Not in Treatment by group |
| Table D.4c | Summary of Present Medical History in Treatment by group |
| Table D.5 | Summary of Patients' Characteristics/Vital Signs at Screening/Baseline by group |
| Table D.6 | Summary of Urine Collection And Storage at Screening/Baseline by group |
| Table D.7 | Summary of Fagerstrom test for nicotine dependence by group |
| Table D.8 | Summary of Step Test at Baseline by group |

| Table number | Efficacy Analyses - Table title |
|---|---|
| Table E.1a | Summary of the Primary End-point. Quit Rate at all visites |
| Table E.1b | Summary of the Primary End-point: Quit Rate at final visit comparison |
| Table E.2 | Summary of the Secondary End-point. Smoking reduction derived from the use of HnB and EC at week 12 |
| Table E.3 | Summary of the Secondary End-point. Adoption rate and adherence to product use at week 12 |
| Table E.4a1 | Summary of the Secondary End-point. mCEQ Questionnaire (scores) by visit |
| Table E.4a2 | Summary of the Secondary End-point. mCEQ Questionnaire. Inferential analysis on the mean changes at final visit from baseline |
| Table E.4b1 | Summary of the Secondary End-point. Smoking Cue Appeal Questionnaire (questions) by visit |
| Table E.4b2 | Summary of the Secondary End-point. Smoking Cue Appeal<br>Questionnaire. Inferential analysis on the mean changes at final visit<br>from baseline |
| Table E.4c2 | Summary of the Secondary End-point. ITUQ Questionnaire. Inferential analysis on the mean changes at final visit from baseline |
| Table E.4d1 | Summary of the Secondary End-point. Risk Perception (PRI-P CC) Questionnaire (scores) by visit |
| Table E.4d2 | Summary of the Secondary End-point. Risk Perception (PRI-P CC). Inferential analysis on the mean changes at final visit from baseline |
| Table E.4e1 | Summary of the Secondary End-point. Risk Perception (PRI-P RRP) Questionnaire (scores) by visit |



Doc code: BIOSTAT.SAP. 02

Pag. 24 of 115

| Table E.4e2 | Summary of the Secondary End-point. Risk Perception (PRI-P RRP) Questionnaire. Inferential analysis on the mean changes at final visit from baseline |
|---|---|
| Table E.4f | Summary of the Secondary End-point. Device delivery by group |
| Table E.5 | Summary of the Secondary Endpoint. Biomarkers of Biological Exposure (BoBE) - eCO (ppm) |
| Table E.6 | Summary of the Secondary Endpoint. EQ-5D questionnaire |
| Table E.7a | Summary of the Secondary Endpoint. Step test by visit |
| Table E.7b | Step test – inferential analysis of VO2MAX |

| Table number | Safety Analyses - Table title |
|--------------|------------------------------------------------------|
| Table \$.1 | Summary of Exent of Exposure and Compliance by group |
| Table \$.2 | Summary of AEs by group |
| Table \$.3 | Summary of Vital Signs by Visit |
| Table S.4 | Summary of End Study Information |

| Listing number | Listing title |
|----------------|-----------------------------------------|
| Listing D.1 | Patients' Disposition |
| Listing D.2 | Eligibility: Inclusion Criteria |
| Listing D.3 | Eligibility: Exclusion Criteria |
| Listing D.4a | Demographic Data |
| Listing D.4b | Smoking Information |
| Listing D.5 | Past and Present Medical History |
| Listing D.6 | Urine collection and Storage |
| Listing D.7 | Fagerstrom test for nicotine dependence |
| Listing D.8 | Step Test |



Doc code: BIOSTAT.SAP. 02

Pag. 25 of 115

| Listing D.9 | Device Consignment |
|--------------|-------------------------------------------|
| Listing D.10 | Product use recording |
| Listing E.1 | EQ-5D |
| Listing E.2 | mCE Questionnaire |
| Listing E.3 | Smoking Cue Appeal Questionnaire |
| Listing E.4 | ITUQ Questionnaire |
| Listing E.5 | Risk Perception (PRI-P CC) Questionnaire |
| Listing E.6 | Risk Perception (PRI-P RRP) Questionnaire |
| Listing S.1 | Extent of Exposure and Study Duration |
| Listing S.2 | Adverse Events |
| Listing S.3 | Vital Signs |



Doc code: BIOSTAT.SAP. 02

Pag. 26 of 115

APPENDIX 2
Mock tables: Tables



Doc code: BIOSTAT.SAP. 02

Pag. 27 of 115

# **BASELINE CHARACTERISTICS**



Doc code: BIOSTAT.SAP. 02

Pag. 28 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.1 Patients Accountability by group Population: All enrolled subjects

| - | 3 | |
|------------------------|--------------|--------------|
| | Group HnB | Group EC |
| Enrolled | XXXX (XX.X%) | XXXX (XX.X%) |
| Screening failures | XXXX (XX.X%) | XXXX (XX.X%) |
| Safety | XXXX (XX.X%) | XXXX (XX.X%) |
| Intention-To-Treat | XXXX (XX.X%) | XXXX (XX.X%) |
| Reason for withdrawal: | | |
| Reason 1 | XX (XX.X%) | XX (XX.X%) |
| Reason 2 | XX (XX.X%) | XX (XX.X%) |
| Reason 3 | XX (XX.X%) | XX (XX.X%) |



Doc code: BIOSTAT.SAP. 02

Pag. 29 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.2a Summary of Demographic and Screening/Baseline Characteristics by group Population: Safety

| | | Group HnB | Group EC |
|----------------------|------------------|------------|------------|
| Age at the time | N | XX | XX |
| of IC Signature Date | N missing | XX | XX |
| | Mean | XX.X | XX.X |
| | Std. deviation | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q1-Q3 | XX.X | XX.X |
| Gender at birth | Male | XX (XX.X%) | XX (XX.X%) |
| | Female | XX (XX.X%) | XX (XX.X%) |
| Education | Primary School | XX (XX.X%) | XX (XX.X%) |
| | Secondary School | XX (XX.X%) | XX (XX.X%) |
| | High School | XX (XX.X%) | XX (XX.X%) |
| | University | XX (XX.X%) | XX (XX.X%) |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>
<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat>
For further information see Listing D.4

Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 30 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.2b Summary of Smoking Information at Screening/Baseline by group (1 of 2) Population: Safety

| | | Group HnB | Group EC | |
|---|---|---|---|---|
| | | N=XXXX | N=XXXX | _ |
| N. cigarettes/die | N<br>N | XX | | XX |
| Screening | N missing<br>Mean | XX.X | | XX.X |
| | Std. deviation Median | XX.X<br>XX.X | | XX.X<br>XX.X |
| | Q1-Q3 | x.x - xx.x | Х | .x - xx.x |
| How long has the subject smoked at least 10 | N<br>N missing | XX<br>XX | | XX<br>XX |
| cigarettes/die? | Mean | XX.X | | XX.X |
| (years) | Std. deviation Median | XX.X<br>XX.X | | XX.X<br>XX.X |
| | Q1-Q3 | X.X - XX.X | Х | .x - xx.x |
| Years of Smoking | N | XX | | XX |
| (years) | N missing | XX<br>XX.X | | XX<br>XX.X |
| | Mean<br>Std. deviation | | | XX.X<br>XX.X |
| | Median | XX.X | | XX.X |
| | Q1-Q3 | x.x - xx.x | X | .x - xx.x |
| N. of quit attempts | N | XX | | XX |
| | N missing | XX | | XX |
| | Mean | XX.X | | XX.X |
| | Std. deviation | | | XX.X |
| | Median | XX.X<br>X.X - XX.X | V | XX.X<br>.X - XX.X |
| | Q1-Q3 | x.x - xx.x | X | .x - xx.x |
| Exhaled breath Carbon | N | XX | | XX |
| monoxide (eCO) Screening | - | XX | | XX |
| (ppm) | Mean | XX.X | | XX.X |
| | Std. deviation | | | XX.X |
| | Median | XX.X | 17 | XX.X |
| | Q1-Q3 | X.X - XX.X | X | .x - xx.x |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>
<Source: [ ]\\Work\_In\_Progress\[ ]\Gestione\_Dati\Dati\_SAS\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat>
For further information see Listing D.5

Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 31 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.2b Summary of Smoking Information at Screening/Baseline by group (2 of 2) Population: Safety

| | | Group HnB<br>N=XXXX | Group EC |
|---|---|---|---|
| Brand of used cigarettes | Brand#1 | XX (XX.X%) | XX (XX.X%) |
| | Brand#2 | XX (XX.X%) | XX (XX.X%) |
| | • • • • • • Brand#n | XX (XX.X%) | XX (XX.X%) |



Doc code: BIOSTAT.SAP. 02

Pag. 32 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Treatment: HnB vs EC

Table D.3 Summary of Past Medical History by group

Population: Safety

| | | Group HnB | Group EC |
|--------------------|-------------------|------------|------------|
| System Organ Class | Preferred Term | N=XXXX | N=XXXX |
| SOC #1 | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| SOC #2 | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| SOC #n | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX
The percentages are computed considering the total of the past medical history abnormalities by group

Coded using MedDRA dictionary (<last available version>)



Doc code: BIOSTAT.SAP. 02

Pag. 33 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.4a Summary of Present Medical History by group

Population: Safety

| ropulation. Salety | | Group HnB | Group EC |
|--------------------|-------------------|------------|------------|
| System Organ Class | Preferred Term | N=XXXX | N=XXXX |
| SOC #1 | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| SOC #2 | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| SOC #n | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati\SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX
The percentages are computed considering the total of the current medical history abnormalities by group
Coded using MedDRA dictionary (<last available version>)



Doc code: BIOSTAT.SAP. 02

Pag. 34 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.4b Summary of Present Medical History not in Treatment by group Population: Safety

| | | Group HnB | Group EC |
|--------------------|-------------------|------------|------------|
| System Organ Class | Preferred Term | N=XXXX | N=XXXX |
| SOC #1 | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| SOC #2 | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| SOC #n | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati\SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX
The percentages are computed considering the total of the current medical history abnormalities by group
Coded using MedDRA dictionary (<last available version>)



Doc code: BIOSTAT.SAP. 02

Pag. 35 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.4c Summary of Present Medical History in Treatment by group

| Population: Safety | | Group HnB | Group EC |
|--------------------|-------------------|------------|------------|
| System Organ Class | Preferred Term | N=XXXX | N=XXXX |
| SOC #1 | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| SOC #2 | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |
| SOC #n | TOTAL | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #1 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #2 | XX (XX.X%) | XX (XX.X%) |
| | PREFERRED TERM #n | XX (XX.X%) | XX (XX.X%) |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX
The percentages are computed considering the total of the current medical history abnormalities by group

Coded using MedDRA dictionary (<last available version>)



Doc code: BIOSTAT.SAP. 02

Pag. 36 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.5 Summary of Patients' Characteristics/Vital Signs at Baseline by group. (1 of n) Population: <Safety/Continuous Quitter>

| Parameter | Statistic | Group HnB | Group EC |
|--------------|----------------|--------------|--------------|
| | | N=XXXX | N=XXXX |
| Parameter #1 | N | XX | XX |
| <um></um> | N missing | XX | XX |
| | Mean | XXX.X | XXX.X |
| | Std. deviation | XX.X | XX.X |
| | Median | XXX.X | XXX.X |
| | Q1-Q3 | XX.X - XXX.X | XX.X - XXX.X |
| Parameter #2 | N | XX | XX |
| <um></um> | N missing | XX | XX |
| | Mean | XXX.X | XXX.X |
| | Std. deviation | XX.X | XX.X |
| | Median | XXX.X | XXX.X |
| | Q1-Q3 | XX.X - XXX.X | XX.X - XXX.X |
| | N | XX | XX |
| <um></um> | N missing | XX | XX |
| | Mean | XXX.X | XXX.X |
| | Std. deviation | XX.X | XX.X |
| | Median | XXX.X | XXX.X |
| | Q1-Q3 | XX.X - XXX.X | XX.X - XXX.X |
| Parameter #n | N | XX | XX |
| <um></um> | N missing | XX | XX |
| | Mean | XXX.X | XXX.X |
| | Std. deviation | XX.X | XX.X |
| | Median | XXX.X | XXX.X |
| | Q1-Q3 | XX.X - XXX.X | XX.X - XXX.X |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>


Doc code: BIOSTAT.SAP. 02

Pag. 37 of 115

Table D.6 Summary of Urine Collection And Storage at Screening/Baseline by group Population: Safety

| | | Group HnB<br>N=XXXX | Group EC |
|---|---|---|---|
| Instruction for urine collection and storage given to the subject | Yes<br>No | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| N. of unire containers<br>Delivered | N<br>N missing<br>Mean<br>Std. deviation<br>Median<br>Q1-Q3 | XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| Has the subject returned the urine to the center? (Baseline) | | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |

<sup>&</sup>lt;File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>
<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX
For further information see Listing X.X



Doc code: BIOSTAT.SAP. 02

Pag. 38 of 115

Table D.7 Summary of Fagerstrom test for nicotine dependence by group Population: Safety

| | | Group HnB | Group EC |
|---|---|---|---|
| | | N=XXXX | N=XXXX |
| Quanto tempo dopo il risveglio fuma la | Entro 5 min | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| prima sigaretta? | Dopo 31-60 min<br>Dopo 60 min | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Trova difficile non fumare nei luoghi dove è vietato? | Si<br>No | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| A quale sigaretta<br>farebbe più fatica a<br>rinunciare? | Alla 1^ del<br>mattino<br>A qualsiasi<br>altra | XX (XX.X%) XX (XX.X%) | XX (XX.X%) XX (XX.X%) |
| Quante sigarette fuma al giorno? | Più di 30<br>21-30<br>11-20<br>10 o meno | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Tende a fumare più<br>spesso nelle prime ore<br>dopo il risveglio che<br>durante il resto del<br>giorno? | Si<br>No | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Fuma anche se è malato<br>e deve rimanere a letto<br>la maggior parte del<br>giorno? | Si<br>No | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |



Doc code: BIOSTAT.SAP. 02

Pag. 39 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table D.8a Summary of Step Test, Step1 to Step 5, at Baseline by group Population: Safety

| | | Group HnB | | Group | p EC |
|--------|----------------|------------|------------|------------|------------|
| | | Heart Rate | Sp02 | Heart Rate | Sp02 |
| Step 1 | N | XX | XX | XX | XX |
| _ | N missing | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | Std. deviation | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Q1-Q3 | X.X - XX.X | X.X - XX.X | X.X - XX.X | X.X - XX.X |
| | N | XX | XX | XX | XX |
| | N missing | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | Std. deviation | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Q1-Q3 | X.X - XX.X | X.X - XX.X | X.X - XX.X | x.x - xx.x |
| Step 5 | N | XX | XX | XX | XX |
| | N missing | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | Std. deviation | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Q1-Q3 | X.X - XX.X | X.X - XX.X | X.X - XX.X | x.x - xx.x |

For further information see Listing X

<sup>&</sup>lt;File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<sup>&</sup>lt;Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 40 of 115

Table D.8b Summary of Step Test, other informations, at Baseline by group Population: Safety

| | | Group | HnB | Group EC | |
|---|---|---|---|---|---|
| | | Heart Rate | Sp02 | Heart Rate | Sp02 |
| Basal Condition | N | XX | XX | XX | XX |
| Recovery Time | N missing | XX | XX | XX | XX |
| (seconds) | Mean | XX.X | XX.X | XX.X | XX.X |
| | Std. deviation | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Q1-Q3 | x.x - xx.x | X.X - XX.X | x.x - xx.x | x.x - xx.x |
| Stop Time | N | XX | : | X | X |
| | N missing | XX | | XX | |
| | Mean | XX. | X | XX.X | |
| | Std. deviation | XX. | X | XX.X | |
| | Median | XX.X | | XX.X | |
| | Q1-Q3 | X.X - XX.X | | X.X - XX.X | |
| VO2MAX | N | XX | | X | X |
| | N missing | XX | • | XX | |
| | Mean | XX. | X | XX.X | |
| | Std. deviation | XX. | X | XX | . X |
| | Median | XX. | X | XX | . X |
| | Q1-Q3 | X.X - | XX.X | X.X - XX.X | |



Doc code: BIOSTAT.SAP. 02

Pag. 41 of 115

# **EFFICACY ENDPOINTS**



Doc code: BIOSTAT.SAP. 02

Pag. 42 of 115

Table E.1a Summary of the Primary End-point. Quit Rate at all visits Population: <Per-Protocol/Intention-To-Treat>

| | | | Group HnB | Group EC |
|-----------|---------|-------|------------|-------------|
| | | | N=XXXX | N=XXXX |
| Quit rate | Visit 1 | N (%) | XXX(XX.X%) | XXX (XX.X%) |
| | Visit 2 | N(%) | XXX(XX.X%) | XXX(XX.X%) |
| | | N(%) | XXX(XX.X%) | XXX(XX.X%) |
| | Visit n | N(%) | XXX(XX.X%) | XXX (XX.X%) |

<sup>&</sup>lt;File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>

<sup>&</sup>lt;Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 43 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.1b Summary of the Primary End-point. Quit Rate at final visit comparison Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC |
|-----------|----------------|------------------------|------------------------|
| | | N=XXXX | N=XXXX |
| Quit Rate | Rate<br>95%CIs | XX.X%<br>[XX.XX,XXX.X] | XX.X%<br>[XX.XX,XXX.X] |

H0: P1-P2 ≤ -Margin H1: P1-P2 > -Margin

Margin=X.XXX

Score (Farrington-Manning)

| Proportion Difference | ASE (F-M) | Z | Pr>Z |
|-----------------------|---------------|--------|--------|
| X.XXXX | X.XXXX | X.XXXX | X.XXXX |
| Noninferiority Limit | 95% Confedent | Limits | |
| X,XXXX | X.XXXX | X.XXXX | |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX
As for the PP population, a "Continuous Quitter" is defined as the subject who did not smoke conventional signrettes from visit 4 to visit 6

For further information see Listing X.X



Doc code: BIOSTAT.SAP. 02

Pag. 44 of 115

Table E.2a Summary of Smoking Reduction derived from the use of HnB and EC at week 12 Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC | p-value |
|---|---|---|---|---|
| | | N=XXXX | N=XXXX | |
| Smoking<br>Reduction | Rate<br>95%CIs | XX.X%<br>[XX.XX,XXX.X] | XX.X%<br>[XX.XX,XXX.X] | X.XXXX |



Doc code: BIOSTAT.SAP. 02

Pag. 45 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.2b Summary of Smoking Reduction derived from the use of HnB and EC according to the Russell Standard Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC | |
|----------------|--------|---------------|---------------|---------|
| Quit timepoint | | N=XXX | N=XXX | p-value |
| Self-reported | Rate | XX.X% | XX.X% | X.XXXX |
| 4 week | 95%CIs | [XX.XX,XXX.X] | [XX.XX,XXX.X] | |
| eCO checked* | Rate | XX.X% | XX.X% | X.XXXX |
| 4 weeks | 95%CIs | [XX.XX,XXX.X] | [XX.XX,XXX.X] | |
| eCO checked* | Rate | XX.X% | XX.X% | X.XXXX |
| 12 weeks | 95%CIs | [XX.XX,XXX.X] | [XX.XX,XXX.X] | |
| eCO checked* | Rate | XX.X% | XX.X% | X.XXXX |
| 24 weeks | 95%CIs | [XX.XX,XXX.X] | [XX.XX,XXX.X] | |
| Lost to FU | Rate | XX.X% | XX.X% | X.XXXX |
| 24 weeks | 95%CIs | [XX.XX,XXX.X] | [XX.XX,XXX.X] | |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>
<Source: [..]\\Work\_In\_Progress\[..]\\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<sup>\*</sup> expired-air 'CO-verified (eCO) 4-week quitter' is the subject that was found to be less than 10ppm in the past 2 weeks The p-value was derived from the XXXX test For further information see Listing X.X



Doc code: BIOSTAT.SAP. 02

Pag. 46 of 115

Table E.3 Summary of Adoption Rate and Adherence to product use at week 12 Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC | p-value |
|---|---|---|---|---|
| | | N=XXXX | N=XXXX | |
| Adoption Rate | Rate<br>95%CIs | XX.X%<br>[XX.XX,XXX.X] | XX.X%<br>[XX.XX,XXX.X] | x.xxxx |



Doc code: BIOSTAT.SAP. 02

Pag. 47 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.4al Summary of the mCE Questionnaire (scores) by visit < Group HnB / Group EC > Population: <Per-Protocol/Intention-To-Treat>

Observed Values at Visit

Changes From Visit 1 to Visits n

| Parameter | | | | | | | | Range | | | | | | | Range |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | N | N miss | Mean | STD | CI 95% | Median | (Q1-Q3) | N | N miss | Mean | STD | CI 95% | Median | (Q1-Q3) |
| Satisfaction | Visit 4 | XX | XX | XX.XX | xx.xx | [XX.XX,XXX.X] | xx.xx | xx.xx - xxx.x | | | | | | | |
| | Visit 5 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | XX.XX - XXX.X | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | XX.XX - XXX.X | | | | | | | |
| | Visit 7 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | xx.xx - xxx.x | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | xx.xx - xxx.x |
| Psychological | Visit 4 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | xx.xx - xxx.x | | | | | | | |
| Reward | Visit 5 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | | | | | | | | |
| | Visit 7 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | xx.xx - xxx.x | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | XX.XX - XXX.X |
| Aversion | Visit 4 | XX | XX | VV VV | xx.xx | [XX.XX,XXX.X] | | xx.xx - xxx.x | | | | | | | |
| 1110131011 | Visit 5 | XX | XX | XX.XX | | [XX.XX,XXX.X] | | XX.XX - XXX.X | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | | [XX.XX,XXX.X] | | | | | | | | | |
| | Visit 7 | XX | XX | | XX.XX | [xx.xx,xxx.x] | | xx.xx - xxx.x | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | XX.XX - XXX.X |
| Enjoyment of | Wigit A | XX | XX | VV VV | xx.xx | [XX.XX,XXX.X] | | xx.xx - xxx.x | | | | | | | |
| Sensation | Visit 5 | XX | XX | | XX.XX | [XX.XX,XXX.X] | | XX.XX - XXX.X | | | | | | | |
| Sensacion | Visit 6 | XX | XX | | XX.XX | [XX.XX,XXX.X] | | | | | | | | | |
| | Visit 7 | XX | XX | | XX.XX | [XX.XX,XXX.X] | | xx.xx - xxx.x | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | XX.XX - XXX.X |
| Craving | Visit 4 | XX | XX | VV VV | XX.XX | [XX.XX,XXX.X] | | xx.xx - xxx.x | | | | | | | |
| Reduction | Visit 5 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | | | | | | | | |
| TICGUCCIOII | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | | | | | | | | |
| | Visit 7 | XX | XX | | XX.XX | [XX.XX,XXX.X] | | xx.xx - xxx.x | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | XX.XX - XXX.X |
| TOTAL | Visit 4 | XX | XX | xx.xx | xx.xx | [XX.XX,XXX.X] | XX.XX | xx.xx - xxx.x | | | | | | | |
| IUIAL | Visit 5 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | | | | | | | | |
| | Visit 6 | XX | XX | | XX.XX | [XX.XX,XXX.X] | | XX.XX - XXX.X | | | | | | | |
| | Visit 7 | XX | XX | | XX.XX | [XX.XX,XXX.X] | | XX.XX - XXX.X | XX | XX | XX XX | XX.XX | [XX.XX,XXX.X] | XX XX | xx.xx - xxx.x |
| | V 1016 / | AA | ΛΛ | ΛΛ.ΛΛ | AA . AA | [^^,^^, | AA.AA | AA.AA AAA.A | AA | ΛΛ | AA.AA | AA.AA | [^^,^^, | AA.AA | nn.nn |



Doc code: BIOSTAT.SAP. 02

Pag. 48 of 115

Table E.4a2 mCE Questionnaire (scores). Inferential analysis on the mean changes at final visit from baseline Population:  $\ensuremath{\mathsf{Per-Protocol}/\mathsf{Intention-To-Treat}}$ 

| | | Group HnB | Group EC | p-value |
|------------------------|------|-----------|----------|---------|
| | | N=XXXX | N=XXXX | |
| Satisfaction | Mean | XX.X | XX.X | X.XXXX |
| Psychological Reward | Mean | XX.X | XX.X | X.XXXX |
| Aversion | Mean | XX.X | XX.X | X.XXXX |
| Enjoyment of Sensation | Mean | XX.X | XX.X | X.XXXX |
| Craving Reduction | Mean | XX.X | xx.x | X.XXXX |
| TOTAL | Mean | XX.X | XX.X | X.XXXX |



Doc code: BIOSTAT.SAP. 02

Pag. 49 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.4b1 Summary of Smoking Cue Appeal Questionnaire by visit. <Question 1 of 8> Population: <Per-Protocol/Intention-To-Treat>

<Question>

| Visit | Score | Group HnB | Group EC |
|---------|-------|------------|-----------|
| | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| | 7 | XX (XX.X%) | XX (XX.X) |
| Visit 5 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| | 7 | XX (XX.X%) | XX (XX.X) |
| Visit 6 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| | 7 | XX (XX.X%) | XX (XX.X) |
| Visit 7 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| | 7 | XX (XX.X%) | XX (XX.X) |

<sup>&</sup>lt;File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

For further information see Listing X.X

<sup>&</sup>lt;Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX

Legend: 1. Estremamente sgradevole ; 2. Molto sgradevole ; 3. Sgradevole ; 4. Né piacevole, né sgradevole ; 5. Piacevole

<sup>6.</sup> Molto piacevole ; 7. Estremamente piacevole



Doc code: BIOSTAT.SAP. 02

Pag. 50 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.4b2 Smoking Cue Appeal Questionnaire. Inferential analysis on the mean changes at final visit from baseline Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC | p-value |
|------------|------|-----------|----------|---------|
| | | N=XXXX | N=XXXX | |
| Question 1 | Mean | XX.X | XX.X | X.XXXX |
| Question 2 | Mean | XX.X | XX.X | X.XXXX |
| | Mean | XX.X | XX.X | X.XXXX |
| Question 8 | Mean | XX.X | XX.X | X.XXXX |
| TOTAL | Mean | XX.X | XX.X | x.xxxx |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat>

For the inferential analysis, the scores were considered as numbers.

The p-value was derived from the XXXX test

For further information see Listing X.X

Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 51 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.4c1 Summary of the ITU Questionnaire by visit. <Question 4 (of questions 4-5-6)> Population: <Per-Protocol/Intention-To-Treat>

#### <Question>

| Visit | Score | Group HnB | Group EC |
|---------|-------|------------|-----------|
| Visit 4 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| | 7 | XX (XX.X%) | XX (XX.X) |
| Visit 5 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| | 7 | XX (XX.X%) | XX (XX.X) |
| Visit 6 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| | 7 | XX (XX.X%) | XX (XX.X) |
| Visit 7 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| | 7 | XX (XX.X%) | XX (XX.X) |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>
<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati\SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX
Legend: 1. Assolutamente falso; 2. Falso; 3. Piuttosto falso; 4. Piuttosto vero; 5. Vero; 6. Molto vero; 7. Verissimo

For further information see Listing X.X



Doc code: BIOSTAT.SAP. 02

Pag. 52 of 115

Table E.4c2 ITU Questionnaire. Inferential analysis on the mean changes at final visit from baseline Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC | p-value |
|------------|------|-----------|----------|---------|
| | | N=XXXX | N=XXXX | |
| Question 4 | Mean | XX.X | XX.X | X.XXXX |
| Question 5 | Mean | XX.X | XX.X | X.XXXX |
| Question 6 | Mean | XX.X | XX.X | X.XXXX |
| TOTAL | Mean | XX.X | xx.x | X.XXXX |



Doc code: BIOSTAT.SAP. 02

Pag. 53 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.4d1 Summary of the Risk Perception (PRI-P CC) Questionnaire by visit. <Question 1 of 18> Population: <Per-Protocol/Intention-To-Treat>

#### <Question>

| Visit | Score | Group HnB | Group EC |
|---------|-------|------------|-----------|
| Visit 4 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 2 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| Visit 5 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| Visit 6 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| Visit 7 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX

Legend: 1. Nessun rischio ; 2. Rischio basso ; 3. Rischio moderato ; 4. Rischio alto ; 5. Rischio molto alto ; 6. Non so

For further information see Listing X.X



Doc code: BIOSTAT.SAP. 02

Pag. 54 of 115

Table E.4d2 Risk Perception (PRI-P CC) Questionnaire. Inferential analysis on the mean changes at final visit from baseline

| | | Group HnB | Group EC | p-value |
|-------------|------|-----------|----------|---------|
| | | N=XXXX | N=XXXX | |
| Question 1 | Mean | XX.X | XX.X | X.XXX |
| Question 2 | Mean | XX.X | XX.X | X.XXX |
| | Mean | XX.X | XX.X | X.XXX |
| Question 18 | Mean | XX.X | XX.X | X.XXX |
| TOTAL | Mean | XX.X | XX.X | X.XXX |

For the inferential analysis, the scores were considered as numbers. Score 6 was not included.



Doc code: BIOSTAT.SAP. 02

Pag. 55 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.4el Summary of the Risk Perception (PRI-P RRP) Questionnaire by visit. <Question 1 of 18> Population: <Per-Protocol/Intention-To-Treat>

<Question>

| Visit | Score | Group HnB | Group EC |
|---------|-------|------------|-----------|
| Visit 4 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| Visit 5 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| Visit 6 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |
| Visit 7 | 1 | XX (XX.X%) | XX (XX.X) |
| | 2 | XX (XX.X%) | XX (XX.X) |
| | 3 | XX (XX.X%) | XX (XX.X) |
| | 4 | XX (XX.X%) | XX (XX.X) |
| | 5 | XX (XX.X%) | XX (XX.X) |
| | 6 | XX (XX.X%) | XX (XX.X) |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX
Legend: 1. Nessun rischio ; 2. Rischio basso ; 3. Rischio moderato ; 4. Rischio alto ; 5. Rischio molto alto ; 6. Non so

For further information see Listing X.X



Doc code: BIOSTAT.SAP. 02

Pag. 56 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.4e2 Risk Perception (PRI-P RRP) Questionnaire. Inferential analysis on the mean changes at final visit from baseline Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC | p-value |
|-------------|------|-----------|----------|---------|
| | | N=XXXX | N=XXXX | |
| Question 1 | Mean | XX.X | XX.X | X.XXXX |
| Question 2 | Mean | XX.X | XX.X | X.XXXX |
| | Mean | XX.X | XX.X | X.XXXX |
| Question 18 | Mean | XX.X | XX.X | X.XXXX |
| TOTAL | Mean | XX.X | XX.X | X.XXXX |

For the inferential analysis, the scores were considered as numbers. Score 6 was not included.



Doc code: BIOSTAT.SAP. 02

Pag. 57 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.4f Summary of Device Delivery by group
Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC |
|---|---|---|---|
| | | N=XXXX | N=XXXX |
| Preferred flavor of chopstick chosen | Heets Amber | XX (XX.X%) | XX (XX.X%) |
| | Heets Yellow | XX (XX.X%) | XX (XX.X%) |
| | Heets Turquoise | XX (XX.X%) | XX (XX.X%) |
| Has the devices been tested and does it works? | Yes | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) |
| Has the subject been trained for the allocated device? | Yes | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat>

For further information see Listing X.X

Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 58 of 115

Table E.5 Summary of the Biomarkers of Biological Exposure (BoBE) - eCO (ppm) Population: <Per-Protocol/Intention-To-Treat>

| | | | | | Observe | d Values at Vis | it | | Changes From Visit 1 to Visits n | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | N | N miss | Mean | STD | CI 95% | Median | Range (Q1-Q3) | N | N miss | Mean | STD | CI 95% | Median | Range (Q1-Q3) |
| Group HnB | Screening | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | xx.xx | (XX.XX - XXX.X) | | | | | | | |
| - | Visit 1 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | |
| | Visit 2 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (xx.xx - xxx.x) | | | | | | | |
| | Visit 3 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | |
| | Visit 4 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | |
| | Visit 5 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | |
| | Follow-up | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) |
| Group EC | Screening | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | |
| | Visit 1 | XX | XX | XX.XX | | [XX.XX,XXX.X] | | (xx.xx - xxx.x) | | | | | | | |
| | Visit 2 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (xx.xx - xxx.x) | | | | | | | |
| | Visit 3 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (xx.xx - xxx.x) | | | | | | | |
| | Visit 4 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (xx.xx - xxx.x) | | | | | | | |
| | Visit 5 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | |
| | Follow-up | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) |
| p-value=X.XXXX | | | | | | | | | | | | | | | |



Doc code: BIOSTAT.SAP. 02

Pag. 59 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.6 Summary of EQ-5D Questionnaire (scores). < Group HnB / Group EC >
Population: <Per-Protocol/Intention-To-Treat/Continuous Quitters>

| | | | Observed Values at Visit | | | | | | | | Changes From Visit 1 to Visits n | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Visit | N | N miss | Mean | STD | CI 95% | Median | min-max | N | N miss | Mean | STD | CI 95% | Median | min-max |
| Mobility | Visit 1 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | | | | | | | |
| (1-5) | Visit 4 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 5 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 6 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 7 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) |
| Self-care | Visit 1 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | | | | | | | |
| (1-5) | Visit 4 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 5 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 6 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 7 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) |
| Health-today | | XX | XX | XX.X | XX.X | [X.X, X.X] | XX.X | (X - X) | | | | | | | |
| (0-100) | Visit 4 | XX | XX | XX.X | XX.X | [X.X, X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 5 | XX | XX | XX.X | XX.X | [X.X, X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 6 | XX | XX | XX.X | XX.X | [X.X, X.X] | XX.X | (X - X) | | | | | | | |
| | Visit 7 | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) | XX | XX | XX.X | XX.X | [X.X , X.X] | XX.X | (X - X) |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat>
For further information see Listing X.X

Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 60 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.7a Summary of Step Test by group < Group HnB / Group EC > Population: <Per-Protocol/Intention-To-Treat>

| | | | Observed Values at Visit | | | | | | | | Changes From Visit 1 to Visit 7 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Visit | N | N miss | Mean | STD | CI 95% | Median | Range (Q1-Q3) | N | N miss | Mean | STD | CI 95% | Median | Range (Q | 1-Q3) |
| Baseline | Visit 1 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | xx.xx | (XX.XX - XXX.X) | | | | | | | | |
| HR | Visit 4 | XX | XX | XX.XX | | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 7 | XX | XX | | XX.XX | [xx.xx,xxx.x] | | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - | XXX.X) |
| SpO2 | Visit 1 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| - | Visit 4 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 7 | XX | XX | | XX.XX | [xx.xx,xxx.x] | | (xx.xx - xxx.x) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - | XXX.X) |
| Step 1 | Visit 1 | XX | XX | | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | | |
| HR | Visit 4 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 7 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - | XXX.X) |
| SpO2 | Visit 1 | XX | XX | XX.XX | | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 4 | XX | XX | XX.XX | | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 7 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - | XXX.X) |
| Recovery | Visit 1 | XX | XX | XX.XX | | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| HR | Visit 4 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | _ | | | |
| | Visit 7 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - | XXX.X) |
| Sp02 | Visit 1 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| - | Visit 4 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 6 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | | |
| | Visit 7 | XX | XX | | XX.XX | [xx.xx,xxx.x] | | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - | XXX.X) |

For further information see Listing X.X

<sup>&</sup>lt;File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<sup>&</sup>lt;Source: [..]\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX
The percentages are calculated on the total of the enrolled patients by group



Doc code: BIOSTAT.SAP. 02

Pag. 61 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table E.7b Summary of Step Test - inferential analysis of VO2MAX Population: <Per-Protocol/Intention-To-Treat>

| | | Group HnB | Group EC |
|--------|----------------|------------|------------|
| VO2MAX | N | XX | XX |
| | N missing | XX | XX |
| | Mean | XX.X | XX.X |
| | Std. deviation | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q1-Q3 | X.X - XX.X | x.x - xx.x |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX

The p-values was derived from the t-test For further information see Listing X



Doc code: BIOSTAT.SAP. 02

Pag. 62 of 115

# **SAFETY ENDPOINTS**



Doc code: BIOSTAT.SAP. 02

Pag. 63 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table S.1 Summary of Extent of Exposure by group

Population: Safety

| | | Group HnB | Group EC |
|----------|----------------|-------------|-------------|
| | | N=XXX | N=XXX |
| Extent | N | XX | XX |
| of | N missing | XX | XX |
| Exposure | Mean | XX.X | XX.X |
| | Std. deviation | XX.X | XX.X |
| | Median | XX.X | XX.X |
| | Q1-Q3 | XX.X - XX.X | XX.X - XX.X |



Doc code: BIOSTAT.SAP. 02

Pag. 64 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table S.2 Summary of Adverse Drug Reactions by group

Population: Safety

| Group HnB | Group EC |
|------------|-------------------------------|
| N=XXX | N=XXX |
| XX (XX.X%) | XX (XX.X%) |
| XX (XX.X%) | XX (XX.X%) |
| XX (XX.X%) | XX (XX.X%) |
| | N=XXX XX (XX.X%) XX (XX.X%) |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>
<Source: [..]\\Work\_In\_Progress\[..]\Gestione\_Dati\Dati\SAS\xxxxx.sas7bdat>

Generated on XXXXXXXXX XX:XX

The percentages are calculated on the total of the enrolled patients by group ADRS classified as Possible/Probably/Definite are considered as Related ADRS For further information see Listing X.X



Doc code: BIOSTAT.SAP. 02

Pag. 65 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy

Protocol: Progetto e-cig vs IQOS

Table S.3 Summary of Vital Signs by group < Group HnB / Group EC >

Population: <Safety/Continuous Quitters>

| | | | | Ob | served 1 | Values at Visit | | | | | Chang | es From | Visit 1 to Visi | ts 6 and | 7 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter<br><unit></unit> | Visit | N | N miss | Mean | STD | CI 95% | Median | Range (Q1-Q3) | N | N miss | Mean | STD | CI 95% | Median | Range (Q1-Q3) |
| parameter #1 | Baseline | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | xx.xx | (XX.XX - XXX.X) | | | | | | | |
| <um></um> | Visit 2 | XX | XX | XX.XX | | [xx.xx,xxx.x] | | (xx.xx - xxx.x) | | | | | | | |
| | Follow-up | XX | XX | XX.XX<br>XX.XX | | [XX.XX,XXX.X]<br>[XX.XX,XXX.X] | | (XX.XX - XXX.X)<br>(XX.XX - XXX.X) | XX | XX<br>XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | [XX.XX,XXX.X]<br>[XX.XX,XXX.X] | XX.XX<br>XX.XX | (XX.XX - XXX.X)<br>(XX.XX - XXX.X) |
| parameter #2 | Baseline | XX | XX | XX.XX | xx.xx | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | |
| <pre>cum&gt;</pre> | Visit 2 | XX | XX | | | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | | | | | | | |
| | | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) |
| | Follow-up | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) |
| parameter #n | Baseline | XX | XX | XX.XX | xx.xx | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | |
| <um></um> | Visit 2 | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | | | | | | | |
| | | XX | XX | XX.XX | | [XX.XX,XXX.X] | | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) |
| | Follow-up | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) | XX | XX | XX.XX | XX.XX | [XX.XX,XXX.X] | XX.XX | (XX.XX - XXX.X) |



Doc code: BIOSTAT.SAP. 02

Pag. 66 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Table S.4 Summary of End of Study Information by group Population: Safety

| | | Group HnB | Group EC |
|---|---|---|---|
| | | N=XXXX | N=XXXX |
| Was the study completed According to the Protocol? | Yes<br>No | XX (XX.X%)<br>XX (XX,X%) | XX (XX.X%)<br>XX (XX.X%) |
| Study duration (days) | N<br>N missing<br>Mean<br>Std. deviation<br>Median<br>Q25-Q75 | XX<br>XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| If no, specify (Reason) | Reason#1 Reason#2 Reason#n | XX (XX.X%)<br>XX (XX.X%)<br> | XX (XX.X%)<br>XX (XX.X%)<br><br>XX (XX.X%) |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>
<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat>

Generated on XXXXXXXXX XX:XX

For further information see Listing X.X



Doc code: BIOSTAT.SAP. 02

Pag. 67 of 115

APPENDIX 3
Mock tables: Listings



Doc code: BIOSTAT.SAP. 02

Pag. 68 of 115

## **BASELINE CHARACTERISTICS**



Doc code: BIOSTAT.SAP. 02

Pag. 69 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing D.1 Patients' Disposition

| Screening<br>Number | Random.<br>Number | Age/Gender | Enroled (Y/N) | Completed (Y/N) |
|---|---|---|---|---|
| xxxxx | xxxxx | XX/XXXX | Х | Х |
| XXXXX | XXXXX | XX/XXXX | X | X |
| XXXXX | XXXXX | XX/XXXX | X | X |
| XXXXX | XXXXX | XX/XXXX | X | X |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>
<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 70 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy

Protocol: Progetto e-cig vs IQOS

Listing D.2 Eligibility: Inclusion Criteria < Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Inclusion<br>Crit. #1 | Inclusion<br>Crit. #2 | Inclusion<br>Crit. #3 | Inclusion<br>Crit. #4 | Inclusion<br>Crit. #5 | Inclusion<br>Crit. #6 |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | XX/XXXX | Х | X | X | X | X | Х |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X | X | X |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

Incl.Crit.#1: Able to comply with study procedures.

Incl.Crit.#2: Male or female healthy smokers aged  $\geq 19$ .

Incl.Crit.#3: Smoking at least 10 cigarettes a day.

Incl.Crit.#4: Smoking for at least one year.

Incl.Crit.#5: Not currently attempting to quit smoking or wishing to do so in the next 30 days (this will be verified at screening by the answer 'NO'' to both questions 'Do you intend to quit in the next 30 days?'' and 'Are you interested in taking part in one of our smoking cessation programs?'').

Incl.Crit.#6: Female smokers not planning to become pregnant are using an acceptable form of contraception.

<Ordered by: Screening Number>

<Stratified by: Group>



Doc code: BIOSTAT.SAP. 02

Pag. 71 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-ciq vs IQOS

Listing D.3 Eligibility: Exclusion Criteria <Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Exclusion<br>Crit. #1 | Exclusion<br>Crit. #2 | Exclusion<br>Crit. #3 | Exclusion<br>Crit. #4 |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | XX/XXXX | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | X |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | Χ |
| XXXXXX | XXXXXX | XX/XXXX | X | X | X | Χ |

<File: [..]\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

Excl.Crit.#1: Use of smokeless tobacco, or any other tobacco products (including e-cigarettes, cigars, chewing tobacco, snus, etc.) within the last 3 months, at baseline and during the whole study;

Excl.Crit.#2: Use of nicotine replacement therapy or other smoking cessation therapies within the last 3 months and at baseline;

Excl.Crit.#3: Self-reported pregnancy, planned pregnancy or breastfeeding;

Excl.Crit.#4: Tobacco industry employees and 1st degree relatives will be excluded in order to safeguard independence of the study.

<Ordered by: Screening Number>

<Stratified by: Group>



Doc code: BIOSTAT.SAP. 02

Pag. 72 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing D.4a Demographic Data < Group HnB / Group EC >

| Screening | Random. | Inf. Cons. | | |
|---|---|---|---|---|
| Number | Number | Date | Age/Gender | Education |
| XXXXXX | XXXXXX | XX/XX/XXXX<br>XX/XX/XXXX | XX/XXXX<br>XX/XXXX | XXXXXXXXXX |
| | | , , | , | |
| XXXXXX | XXXXXX | XX/XX/XXXX | XX/XXXX | XXXXXXXXXX |
| XXXXXX | XXXXXX | XX/XX/XXXX | XX/XXXX | XXXXXXXXX |
| XXXXXX | XXXXXX | XX/XX/XXXX | XX/XXXX | XXXXXXXXXX |
| XXXXXX | XXXXXX | XX/XX/XXXX | XX/XXXX | XXXXXXXXX |
| XXXXXX | XXXXXX | XX/XX/XXXX | XX/XXXX | XXXXXXXXXX |
| XXXXXX | XXXXXX | XX/XX/XXXX | XX/XXXX | XXXXXXXXX |
| XXXXXX | XXXXXX | XX/XX/XXXX | XX/XXXX | XXXXXXXXXX |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>

<Stratified by: Group>


Doc code: BIOSTAT.SAP. 02

Pag. 73 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy

Protocol: Progetto e-cig vs IQOS

Listing D.4b Smoking information < Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | How long smoked at least<br>10 cigarettes/die (years) | Brand of used cigarettes | Years of smoking | Number of quit attempts | Visit | Number of cigarette/die | Exhaled breath<br>Carbon monoxide |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XX/XXXX | XX | XXXXXXXXX | XX | XX | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| XXXXXX | XXXXXX | XX/XXXX | XX | XXXXXXXXX | XX | XX | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| XXXXXX | XXXXXX | XX/XXXX | XX | XXXXXXXXX | XX | XX | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |
| | | | | | | | XXXXXX | XX | XXX |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 74 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing D.5 Past and Present Medical History < Group HnB  $\prime$  Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Date of<br>Visit | Description | Date of<br>Onset | Date<br>Resolved | Ongoing<br>(Y/N) | Comment |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | xxxxx | XX/XXXX | XX/XX/XXXX | xxxxxxxx | XX/XX/XXXX | XX/XX/XXXX | X | XXXXXXXXX |
| XXXXXX | XXXXXX | XX/XXXX | XX/XX/XXXX | XXXXXXXXX | XX/XX/XXXX | XX/XX/XXXX | X | XXXXXXXXX |



Doc code: BIOSTAT.SAP. 02

Pag. 75 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing D.6 Urine Collection and Storage < Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Sex | Instruction given to the subject? | No. of urine<br>Containers delivered | Visit | Has the subject returned the urine to the center? |
|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XX.X/XXXX | XXX | XXX | XXXXXXX | 7777 |
| | | | | 373737 | XXXXXXX | XXX |
| | | | | XXX | XXXXXXX | |
| | | | | | XXXXXXX | XXX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXX | XXX | XXXXXXX | |
| | | | | | XXXXXXX | XXX |
| | | | | XXX | XXXXXXX | |
| | | | | | XXXXXXX | XXX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXX | XXX | XXXXXXX | |
| | | | | | XXXXXXX | XXX |
| | | | | XXX | XXXXXXX | |
| | | | | | XXXXXXX | XXX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXX | XXX | XXXXXXX | |
| | | | | | XXXXXXX | XXX |
| | | | | XXX | XXXXXXX | 22221 |
| | | | | 71111 | XXXXXXX | XXX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXX | XXX | XXXXXXX | |
| | | | | | XXXXXXX | XXX |
| | | | | XXX | XXXXXXX | |
| | | | | | XXXXXXX | XXX |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 76 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IOOS

Listing D.7 Fagerstrom test for nicotine dependance < Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Visit | Age/Gender | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXXXXX | XX/XXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |

\_\_\_\_\_

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

- Q1: Quanto tempo dopo il risveglio fuma la prima sigaretta?
- Q2: Trova difficile non fumare nei luoghi dove è vietato?
- Q3: A quale sigaretta farebbe più fatica a rinunciare?
- Q4: Quante sigarette fuma al giorno?
- Q5: Tende a fumare più spesso nelle prime ore dopo il risveglio che durante il resto del giorno?
- Q6: Fuma anche se è malato e deve rimanere a letto la maggior parte del giorno?

<Ordered by: Screening Number>

<sup>&</sup>lt;File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>



Doc code: BIOSTAT.SAP. 02

Pag. 77 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy

Protocol: Progetto e-cig vs IQOS

Listing D.8 Step Test < Group HnB / Group EC >

| Screening | Ranom. | | | Basal | e | Step | 1 | Step | 2 | Step | 3 | Step | 4 | Step | 5 | Recove | ery | Stop | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Number | Age/Gender | Visit | HR | Sp02 | HR | Sp02 | HR | Sp02 | HR | Sp02 | HR | Sp02 | HR | Sp02 | HR | Sp02 | Time | V02MAX |
| XXXXXX | xxxxxx | XX.X/XXXX | xxxxxxx | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| ΛΛΛΛΛΛ | ΛΛΛΛΛΛ | ΛΛ•Λ/ΛΛΛΛ | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | *************************************** | | | | | | | | | | | | | | | ****** | |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| ΛΛΛΛΛΛ | ΛΛΛΛΛΛ | ΛΛ•Λ/ ΛΛΛΛ | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | | XX.X | XX.X | | XX.X | | | XX.X | | XX.X | XX.X | XX.X | XX.X | XX.X | | | |
| | | | XXXXXXX | AA.A | XX.X | XX.X | AA.A | XX.X | XX.X | XX.X | XX.X | XX.X | AA.A | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |
| | | | XXXXXXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XXXX | XX.XX |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 78 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy

Protocol: Progetto e-cig vs IQOS

Listing D.9 Device consignment < Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Visit | Has the device been tested and does it work? | Has the subject been trained for the allocated device? | <pre><see> footnote&gt;</see></pre> | <see<br>footnote&gt;</see<br> |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XX/XXXX | XXXXXX | XXX | XXXXXXXXXX | XXXXX | XXXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXX | XXXXX | XXXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXX | XXXXX | XXXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXX | XXXXX | XXXXXXXXX |
| XXXXXX | XXXXXX | XX/XXXX | XXXXXX | XXX | xxxxxxxxxx | XXXXX | XXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXX | XXXXX | XXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXXX | XXXXX | XXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXX | XXXXX | XXXXXXXXX |
| XXXXXX | XXXXXX | XX/XXXX | XXXXXX | XXX | xxxxxxxxxx | XXXXX | XXXXXXXXX |
| | | , | XXXXXX | XXX | XXXXXXXXXXX | XXXXX | XXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXXX | XXXXX | XXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXX | XXXXX | XXXXXXXXX |
| XXXXXX | XXXXXX | XX/XXXX | XXXXXX | XXX | xxxxxxxxxx | XXXXX | XXXXXXXXX |
| | | , | XXXXXX | XXX | XXXXXXXXXXX | XXXXX | XXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXXX | XXXXX | XXXXXXXXX |
| | | | XXXXXX | XXX | XXXXXXXXXX | XXXXX | XXXXXXXXX |

<File: [..]\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>

<Stratified by: Group>

<No. of sticks delivered - Preferred flavor@of heatstick / Quantity in mg/ml of e-liquid bottles - Preferred flavor@of e-liquid>



Doc code: BIOSTAT.SAP. 02

Pag. 79 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing D.10 Device supply and accountability < Group HnB  $\prime$  Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Visit | <see footnote=""></see> |
|---|---|---|---|---|
| ××××× | XXXXXX | XX/XXXX | xxxxxxx | XXX |
| ΛΛΛΛΛ | ΛΛΛΛΛΛ | ΛΛ/ ΛΛΛΛ | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| XXXXXX | XXXXXX | XX/XXXX | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| XXXXXX | XXXXXX | XX/XXXX | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| XXXXXX | XXXXXX | XX/XXXX | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |
| | | | XXXXXXX | XXX |

<sup>&</sup>lt;File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<sup>&</sup>lt;Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<sup>&</sup>lt;Ordered by: Screening Number>

<sup>&</sup>lt;Stratified by: Group>

<sup>&</sup>lt; Average sticks consumed per day / No. of empty e-liquid refill bottles returned>



Doc code: BIOSTAT.SAP. 02

Pag. 80 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing D.11 Product use recording < Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Q1 | If yes, specify type and amount of daily use | Q2 | If yes, average<br><sticks consumed="" e-liquid="" in="" ml=""> per day</sticks> |
|---|---|---|---|---|---|---|
| XXXXXX | xxxxxx | XX/XXXX | XXX | xxxxxxxxxxxxxxxxx | XXX | XXXXXXXXX |
| XXXXXX | XXXXXX | XX/XXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | xxxxxxxxx |
| XXXXXX | XXXXXX | XX/XXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | xxxxxxxxx |
| XXXXXX | XXXXXX | XX/XXXX | XXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX | xxxxxxxxx |
| XXXXXX | XXXXXX | XX/XXXX | XXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX | xxxxxxxxx |
| XXXXXX | XXXXXX | XX/XXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | xxxxxxxxx |
| XXXXXX | XXXXXX | XX/XXXX | XXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX | xxxxxxxxx |
| XXXXXX | XXXXXX | XX/XXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | xxxxxxxxx |
| XXXXXX | XXXXXX | XX/XXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | xxxxxxxxx |
| XXXXXX | XXXXXX | XX/XXXX | XXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX | xxxxxxxxx |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

Q1: Did the subject use different RRP or other anti-smoking products during the last three months?

Q2: If no, are you using the products delivered by this study?

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 81 of 115

# **EFFICACY DATA**



Doc code: BIOSTAT.SAP. 02

Pag. 82 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing E.1 EQ-5D <Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Visit | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | X | X | X | X | X | XXX |
| | | | XXXXXXX | X | X | X | X | X | XXX |
| | | | XXXXXXX | X | X | X | X | X | XXX |
| | | | XXXXXXX | X | X | Χ | X | X | XXX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | X | Х | Х | Х | Х | XXX |
| | | | XXXXXXX | X | X | X | X | X | XXX |
| | | | XXXXXXX | X | X | X | X | X | XXX |
| | | | XXXXXXX | X | Χ | Χ | Χ | Χ | XXX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Х | Х | Х | Х | XXX |
| | | | XXXXXXX | X | X | X | X | X | XXX |
| | | | XXXXXXX | X | X | X | X | X | XXX |
| | | | XXXXXXX | X | Χ | Χ | Χ | Χ | XXX |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | X | Х | X | X | XXX |
| | | | XXXXXXX | Χ | X | X | X | X | XXX |
| | | | XXXXXXX | Χ | X | X | X | X | XXX |
| | | | XXXXXXX | X | Χ | Χ | Χ | Χ | XXX |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 83 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing E.2 MCEQ <Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Visit | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 | Q9 | Q10 | Q11 | Q12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | X | X | X | X | X | X | X | X | X | X | Χ | X |
| | | | XXXXXXX | X | X | X | X | X | X | X | X | X | X | X | X |
| | | | XXXXXXX | X | X | X | X | X | X | X | X | X | X | X | Χ |
| | | | XXXXXXX | Χ | X | X | Χ | X | Χ | Χ | Χ | X | X | X | X |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | X | X | X | X | Χ | Χ | Х | X | Х | X | X |
| | | | XXXXXXX | X | Χ | Χ | Χ | Χ | X | Χ | Χ | Χ | X | Χ | Χ |
| | | | XXXXXXX | X | X | X | Χ | X | X | Χ | X | X | X | Χ | X |
| | | | XXXXXXX | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | X | X | Х | X | Х | Х | Х | Х | X | X | X |
| | | | XXXXXXX | X | X | X | Χ | X | X | Χ | X | Χ | X | Χ | Χ |
| | | | XXXXXXX | X | X | X | Χ | X | X | Χ | X | Χ | X | Χ | X |
| | | | XXXXXXX | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Х | Х | X | Х | X | Χ | Х | Х | X | Х | X |
| | | | XXXXXXX | X | X | X | Χ | X | Χ | X | X | X | X | Χ | X |
| | | | XXXXXXX | X | X | X | Χ | X | X | X | X | X | X | Χ | X |
| | | | XXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 84 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing E.3 Smoking cue appeal <Group HnB / Group EC >

| Screening<br>Number | Random.<br>Number | Age/Gender | Visit | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXXXXX | Χ | X | X | X | X | X | X | Χ |
| | | | XXXXXXX | X | X | X | X | X | X | Χ | X |
| | | | XXXXXXX | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | X | Х | Х | X | X | X | X | Х |
| | | | XXXXXXX | Χ | X | X | X | X | X | X | X |
| | | | XXXXXXX | Χ | Х | Х | Х | Х | X | X | Х |
| | | | XXXXXXX | X | X | X | X | X | X | X | Χ |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Х | Х | X | X | Х | Х | Х |
| | | | XXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXXXXX | X | X | X | X | X | X | X | Х |
| | | | XXXXXXX | X | X | X | X | X | X | X | X |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Х | Х | Х | Х | Х | X | Х |
| | | | XXXXXXX | X | X | X | X | X | X | X | X |
| | | | XXXXXXX | Χ | Х | Х | Х | Х | X | X | X |
| | | | XXXXXXX | X | X | X | X | X | X | X | X |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 85 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing E.4 ITUQ <Group HnB / Group EC >

| Screening | Random. | | | | | |
|-----------|---------|------------|---------|----|----|----|
| Number | Number | Age/Gender | Visit | Q4 | Q5 | Q6 |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | X | X | X |
| | | | XXXXXXX | X | Χ | Χ |
| | | | XXXXXXX | X | X | X |
| | | | XXXXXXX | Χ | Χ | Χ |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | X | Х |
| | | | XXXXXXX | X | X | X |
| | | | XXXXXXX | X | X | X |
| | | | XXXXXXX | Χ | X | Χ |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Χ | Χ |
| | | | XXXXXXX | X | X | X |
| | | | XXXXXXX | X | X | X |
| | | | XXXXXXX | Χ | Χ | Χ |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Χ | Χ |
| | | | XXXXXXX | X | X | X |
| | | | XXXXXXX | Χ | X | X |
| | | | XXXXXXX | Χ | X | Χ |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 86 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy

Protocol: Progetto e-cig vs IQOS

Listing E.5 Risk perception CC <Group HnB / Group EC >

| Screening | Random. | | | Scr | een 1 | /3 | | | | Scr | een 2 | /3 | | | | Scr | een 3 | /3 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Number | Age/Gender | Visit | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 |
| XXXXXX | XXXXXX | XX.X/XXXX | xxxxxxx | Х | X | Х | X | X | Х | X | X | Х | X | X | Х | Х | X | X | X | X | Х |
| ΛΛΛΛΛΛ | ΛΛΛΛΛΛ | ΛΛ•Λ/ ΛΛΛΛ | XXXXXXX | Х | | X | X | Х | X | X | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | X |
| | | | | | X | | | | | | | | | | | | | | | | |
| | | | XXXXXXX | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | | XXXXXXX | Х | Χ | Χ | X | Χ | Χ | Х | X | Х | Χ | Х | Х | Χ | Χ | Х | Х | Х | Χ |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | | | XXXXXXX | X | X | X | X | X | X | X | X | Χ | X | X | X | X | Χ | X | X | X | Χ |
| | | | XXXXXXX | Х | X | X | X | Χ | X | X | X | X | X | X | X | Χ | X | Х | Х | Х | Х |
| | | | XXXXXXX | Х | Χ | Χ | Х | Х | Χ | Χ | Х | Χ | Χ | Χ | Χ | Х | Χ | Х | Х | Х | Х |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | ********* | *************************************** | XXXXXXX | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Х |
| | | | XXXXXXX | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | | | | | | | | | | | | | Х | | | | | | | |
| | | | XXXXXXX | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | Χ | Χ | Χ | X | X | X | Х |
| XXXXXX | XXXXXX | XX.X/XXXX | XXXXXXX | Х | Χ | Χ | Χ | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | | | XXXXXXX | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | | XXXXXXX | Х | X | X | X | Χ | X | X | X | X | X | X | X | Χ | X | Х | Х | Х | Х |
| | | | XXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 87 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy

Protocol: Progetto e-cig vs IQOS

Listing E.6 Risk perception RRP <Group HnB / Group EC >

| Random. | | | Scr | een 1. | /3 | | | | Scr | een 2 | /3 | | | | Scr | een 3. | /3 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Age/Gender | Visit | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 |
| VVVVV | VV V/VVV | | ~ | | ~ | v | | | | | | | | ~ | | | | | | X |
| ΛΛΛΛΛΛ | ΛΛ•Λ/ ΛΛΛΛ | | | | | | | | | | | | | | | | | | | X |
| | | | | | | | | | | | | | | | | | | | | X |
| | | XXXXXXX | X | Χ | Χ | Χ | Χ | Χ | Λ | Λ | Χ | X | X | X | Χ | Χ | Λ | Λ | Λ | Х |
| XXXXXX | XX.X/XXXX | XXXXXXX | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | | XXXXXXX | X | X | X | X | Χ | Χ | X | Χ | Χ | X | X | X | Χ | X | X | X | X | X |
| | | XXXXXXX | X | X | Х | X | X | X | X | X | Χ | Х | Х | Х | X | Χ | X | Х | X | X |
| | | XXXXXXX | Х | Χ | Χ | Χ | Χ | Χ | Χ | X | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Х |
| XXXXXX | xx.x/xxxx | XXXXXXX | Х | Х | X | Х | Х | Х | Х | X | Х | Х | Х | Х | X | Х | X | X | X | Х |
| | | | | | | | | | | | | | | | | | | | | Х |
| | | | | | | | | | | | | | | | | | | | | Х |
| | | | | | | | | | | | | | | | | | | | | X |
| | | XXXXXXX | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ |
| XXXXXX | XX.X/XXXX | XXXXXXX | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х |
| | | XXXXXXX | X | X | X | X | X | X | X | Χ | Χ | X | X | X | Χ | X | X | X | X | X |
| | | XXXXXXX | X | X | X | X | Χ | Χ | X | Χ | Χ | X | X | X | Χ | X | X | X | X | X |
| | | XXXXXXX | Х | X | X | X | Χ | X | X | X | X | X | X | X | X | X | Х | Х | Х | X |
| | Number XXXXXX XXXXXX | Number Age/Gender XXXXXX XX.X/XXXX XXXXXX XX.X/XXXX XXXXXX XX.X/XXXX | Number Age/Gender Visit XXXXXX XX.X/XXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXX XX.X/XXXX XXXXXXX XXXXXX XXXXXXX XXXXXXX XXXXXX XXXXXXX XXXXXXX XXXXXX XXXXXXX XXXXXXX XXXXXX XXXXXXX XXXXXXX XXXXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXXX XXXXXXX XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXX XXXXXXXXXXXX< | Number Age/Gender Visit Q1 XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXXX XXXXXXXXXXXX XXXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Number Age/Gender Visit Q1 Q2 XXXXXX XX.X/XXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXXXX XXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Number Age/Gender Visit Q1 Q2 Q3 XXXXXXX XX.X/XXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Number Age/Gender Visit Q1 Q2 Q3 Q4 XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 XXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXXX XXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 XXXXXXX XX.XXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 XXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXX XXXXXXXXXXX XXXXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX <t< td=""><td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXX<td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX</td><td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 XXXXXXX XXXXXXXX XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX</td><td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X</td><td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X</td></td></t<> <td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X &lt;</td> <td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 XXXXXXX X X X X X X X X X X X X X X X X X X X X X X<td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q5 Q6 Q1 Q2 Q3 Q4 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X &lt;</td><td> Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q5 Q5 Q5 Q5 Q5</td></td> | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXX XXXXXXXXXX XXXXXXXXXX <td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX</td> <td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 XXXXXXX XXXXXXXX XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX</td> <td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X</td> <td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X</td> | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 XXXXXXX XXXXXXXX XXXXXXXX | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 XXXXXXX XXXXXXXX XXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXX | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X < | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 XXXXXXX X X X X X X X X X X X X X X X X X X X X X X <td>Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q5 Q6 Q1 Q2 Q3 Q4 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X &lt;</td> <td> Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q5 Q5 Q5 Q5 Q5</td> | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q5 Q6 Q1 Q2 Q3 Q4 XXXXXXX XXXXXXXX X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X < | Number Age/Gender Visit Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q6 Q1 Q2 Q3 Q4 Q5 Q5 Q5 Q5 Q5 Q5 Q5 |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.sas7bdat> Generated on XXXXXXXXX XX:XX

<Ordered by: Screening Number>



Doc code: BIOSTAT.SAP. 02

Pag. 88 of 115

# **SAFETY DATA**



Doc code: BIOSTAT.SAP. 02

Pag. 89 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing S.1 Extent of Exposure and Study Duration <Group HnB  $\prime$  Group EC >

| Screening<br>Number | Random.<br>Number | Age/Sex | Visit | Start<br>Date | End<br>Date | Days of<br>Exposure |
|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | XX.X/XXXX | XX | XX/XX/XXXX | XX/XX/XXXX | XXX |
| XXXXXX | XXXXXX | XX.X/XXXX | XX | XX/XX/XXXX | XX/XX/XXXX | XXX |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\\Work\_In\_Progress\[..]\Gestiona Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 90 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-ciq vs IQOS

Listing S.2 Adverse Events <Group HnB / Group EC >

| Screen. | Random. | | N. | AE | If other | AE | Is the AE | | If Death | If death | If hospital | ization | | If recovery, | Relations | Action |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Number | Age/Sex | AE | Description | specify | Severity | Serious? | If Serious | Specify date | autopsy? | Start Date | End Date | Outcome | recovery date | with products? | Taken |
| XXXXXX | XXXXXX | x.x/xxxx | XX | XXXXXXXXX | xxxxxxx | XXX | XXX | xxxxxxxxx | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | xxxxxxx | XX/XX/XXXX | XXX | xxxxxxx |
| XXXXXX | xxxxxx | X.X/XXXX | XX | xxxxxxxxx | xxxxxxxx | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | xxxxxxx | XX/XX/XXXX | XXX | XXXXXXX |
| XXXXXX | xxxxxx | x.x/xxxx | XX | XXXXXXXXX | xxxxxxx | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | xxxxxxx | XX/XX/XXXX | XXX | XXXXXXX |
| XXXXXX | XXXXXX | X.X/XXXX | XX | XXXXXXXXX | xxxxxxx | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | xxxxxxx | XX/XX/XXXX | XXX | XXXXXXX |
| XXXXXX | XXXXXX | X.X/XXXX | XX | XXXXXXXXX | xxxxxxx | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | xxxxxxx | XX/XX/XXXX | XXX | XXXXXXX |
| XXXXXX | XXXXXX | X.X/XXXX | XX | XXXXXXXXX | XXXXXXX | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | XXXXXXX | XX/XX/XXXX | XXX | XXXXXXX |
| XXXXXX | XXXXXX | X.X/XXXX | XX | XXXXXXXXX | xxxxxxx | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | xxxxxxx | XX/XX/XXXX | XXX | XXXXXXX |
| XXXXXX | XXXXXX | X.X/XXXX | XX | XXXXXXXXX | xxxxxxx | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | xxxxxxx | XX/XX/XXXX | XXX | XXXXXXX |
| XXXXXX | XXXXXX | X.X/XXXX | XX | XXXXXXXXX | XXXXXXXX | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | XXXXXXX | XX/XX/XXXX | XXX | XXXXXXX |
| XXXXXX | XXXXXX | X.X/XXXX | XX | XXXXXXXXX | XXXXXXXX | XXX | XXX | XXXXXXXXX | XX/XX/XXXX | XXX | XX/XX/XXXX | XX/XX/XXXX | XXXXXXX | XX/XX/XXXX | XXX | XXXXXXX |

<File: [..]\\Work In Progress\[..]\Statistica\Programmi\xxxxx.sas>

<Source: [..]\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX

AE Severity: 0=Mild; 1=Moderate; 2=Severe

AE Serious: 0=Death; 1=Life threatening; 2=Hospitalization or prolonged hospitalization; 3=Permanent significant disability

4=Congenital anomaly/birth deficit; 5=Medical important event

Outcome: 1=Recovered without Sequelae; 2=Recovered with Sequelae; 3=Ongoing; 4=Persisting; 5=Unknown

Relationship: 0=Not Related; 1=Unlikely; 2=Possible; 1=Probably; 2=Definitive

Action Taken: 0=No action taken; 1=Study product dosage adjusted; 2=Study product temporarily interrupted



Doc code: BIOSTAT.SAP. 02

Pag. 91 of 115

Sponsor: Center for Tobacco Research, Cessation and Prevention, Via S. Sofia 78, 95123, Catania (CT) - Italy Protocol: Progetto e-cig vs IQOS

Listing S.3 Vital Signs <Group HnB / Group EC >

| Screening | | Ago/Condo | 77: 0: + | Date of | Parameter #1 | Parameter #2 | | Parameter #n |
|---|---|---|---|---|---|---|---|---|
| Number | Number | Age/Gender | Visit | Visit | <u.m.></u.m.> | <u.m.></u.m.> | | <u.m.></u.m.> |
| XXXXXX | XXXXXX | XX.X/XXXX | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| 212121212121 | 212121212121 | 2121 • 21 / 21212121 | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| | | | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| | | | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| | | | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| XXXXXX | XXXXXX | XX.X/XXXX | XX | xx/xx/xxxx | XXX.X | XXX.X | XXX.X | XXX.X |
| | | | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| XXXXXX | XXXXXX | XX.X/XXXX | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| | | | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| XXXXXX | XXXXXX | XX.X/XXXX | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| | | | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX.X |
| | | | XX | XX/XX/XXXX | XXX.X | XXX.X | XXX.X | XXX |

<File: [..]\\Work\_In\_Progress\[..]\Statistica\Programmi\xxxxx.sas>

<sup>&</sup>lt;Source: [..]\Work In Progress\[..]\Gestione Dati\Dati SAS\xxxxx.satd7sas> Generated on XXXXXXXXX XX:XX



Doc code: BIOSTAT.SAP. 02

Pag. 92 of 115

APPENDIX 4
Flow Chart



Doc code: BIOSTAT.SAP. 02

Pag. 93 of 115

| | V0<br>screening | V1<br>baseline | V2 | V3 | V4 | V5 | V6 | V7<br>follow-up |
|---|---|---|---|---|---|---|---|---|
| Assessment | | ≤ 7 days<br>after V0 | 1 week<br>after visit<br>1 | 2 weeks<br>after visit<br>1 | 4 weeks<br>after visit<br>1 | 8 weeks<br>after visit<br>1 | 12 weeks<br>after visit<br>1 | 24 weeks<br>after visit<br>1 |
| | | | +/-3 days | +/-3 days | +/-3 days | +/-7 days | +/-7 days | +/-7 days |
| Medical/smoking/vaping/new generation product use history | Х | | | | | | | Х |
| Instructions for urine collection and storage; delivery of containers | Х | | | Х | | | | |
| Eligibility criteria verification and confirmation | Х | | | | | | | |
| Informed consent | Х | | | | | | | |
| Vital Signs (BP, HR) | | Χ | Х | Χ | Х | Х | Χ | Х |
| Weight and Height | | Χ | | | | | Χ | Х |
| Urine sample pick up | | Χ | | | Χ | | | |
| Randomization | | Χ | | | | | | |
| Training for the allocated device (from 30min to 2 hours) | | Х | | | | | | |
| Device delivery (included 1 week supply heatsticks for iQOS or eliquid for JustFog) | | Х | | | | | | |
| Providing 1 week supply of heatsticks for iQOS or eliquid for JustFog | | | Х | | | | | |
| Providing 2 weeks supply of heatsticks for iQOS or eliquid for JustFog | | | | Х | | | | |



Doc code: BIOSTAT.SAP. 02

Pag. 94 of 115

| Providing 4 weeks supply of heatsticks for iQOS or eliquid for JustFog | | | | x | x | | |
|---|---|---|---|---|---|---|---|
| Smoking consumption/abstinence/reduction | Х | Х | Х | Х | Х | Х | Х |
| recording through subject selfreporting | | | | | | | |
| Device and supply accountability (collection of empty e-liquid refill bottles and used heathsticks; eventual substitution of malfunctioning | | Х | х | х | х | х | х |
| devices) | | | | | | | |
| mCEQ | | | | Х | Χ | Χ | Х |
| Smoking Cue Appeal (8 items) | | | | Х | Х | Х | Х |
| ITUQ – items 4-6 | | | | Х | Х | Х | Х |
| Risk perception (PRI-P CC e PRIP RRP) | | | | Х | Χ | Χ | Х |
| EQ-5D | X | | | Χ | Χ | Χ | Х |
| eCO | Х | Χ | Х | X | Χ | Χ | Х |
| Step test | X | | | Х | | Χ | Х |
| Safety and product reliability onitoring reporting | Х | Х | Х | Х | Х | Х | Х |



Doc code: BIOSTAT.SAP. 02

Pag. 95 of 115

APPENDIX 5 DRM Minute



Doc code: BIOSTAT.SAP. 02

Pag. 96 of 115

| <b>Titolo del Protocollo</b> : A 12-weeks open label, non-inferiority trial comparing HnB products vs ECs in terms of efficacy and adoption rates, acceptability, tolerability, and tobacco harm reduction in healthy smokers, not motivated to quit. | Versione: 1.0 26 Settembre 2017 |
|---|---|
| Prodotto: Sigaretta elettronica/HnB (Heat-not-Burn) | Sponsor: AOU Policlinico Vittorio<br>Emanuele - University of Catania<br>Centro per la cura e la prevenzione del<br>tabagismo |
| Contatti:Pasquale Caponnetto - AOU Policlinico Vittorio Emanuele University of Catania Email: p.caponnetto@unict.it - Phone number: (+39) 095.3781537 | |

| REDATTORE | | | |
|---|---|---|---|
| Nome | Qualifica | Data | Firma |
| Maurizio<br>Ceracchi | Statistico<br>Fullcro | 30/06/2020 | Marin Sent. |



Doc code: BIOSTAT.SAP. 02

Pag. 97 of 115

| PARTECIPANTI<br>Nome | | | |
|---|---|---|---|
| Riccardo | Qualifica | Data | Firma |
| Polosa | Direttore | ON 10742020 | Ruc |
| Pasquale<br>Caponnetto | Co-sperimentatore | 0167-12020 | MIGH |
| Fabio<br>Cibella | Consulente Statistico | 01/07/2020 | Feballe |
| Caruso<br>Massimo | Responsabile<br>Laboratorio | 01/07/2020 | Donlus Bus |
| Marilena<br>Maglia | Sub-sperimentatore | 01/07/2020 | MGModia |
| Rosalia<br>Emma | Co-responasabile<br>laboratorio | 01/07/2020 | Roslie Emm |
| /alentina<br>Granelli | Project<br>Manager<br>Fullcro | | |
| drian<br>hallvari | Data<br>Manager<br>Fullcro | | I I I I |

| NON PARTECIPANTI Nome | Qualifica | Data | Firma |
|---|---|---|---|
| Maria | Sperimentatore<br>Principale<br>stra borta annuare po | 01/07/2020 | Sun Jeen |
| alia quale si co<br>gaitto <sup>laurea</sup> .<br>Daujeja | llegheranno anche gli<br>Wauadet<br>Luoject | studenti the dovra | n 10 affrontare l'esame d |



Doc code: BIOSTAT.SAP. 02

Pag. 98 of 115

| PARTECIPANTI | | | |
|---|---|---|---|
| Nome | Qualifica | Data | Firma |
| Riccardo<br>Polosa | Direttore | | |
| Pasquale<br>Caponnetto | Co-sperimentatore | | |
| Fabio<br>Cibella | Consulente Statistico | | |
| Caruso<br>Massimo | Responsabile<br>Laboratorio | | |
| Marilena<br>Maglia | Sub-sperimentatore | | |
| Rosalia<br>Emma | Co-responasabile<br>laboratorio | | |
| Valentina<br>Granelli | Project<br>Manager<br>Fullcro | 01/07/2020 | illemay animold |
| Adrian<br>Shallvari | Data<br>Manager<br>Fullcro | 01/07/2020 | Atz. |



Doc code: BIOSTAT.SAP. 02

Pag. 99 of 115

# STORIA DELLE VERSIONI

| Versione | Data | Descrizione dei cambiamenti |
|---|---|---|
| Draft 0.1 | 12 Giugno 2020 | Prima versione per la revisione del Team |
| Draft 0.2 | 23 Giugno 2020 | Nuova versione successiva ad una call di chiarimento dopo il |
| | | DRM |
| Finale 1.0 | 08 Luglio 2020 | Versione finale dopo la revisione del team |

# INDICE

| 1 | INTRODUZIONE |
|-----|---------------------------------------------------------------------|
| 2 | ARGOMENTI IN AGENDA |
| 2.1 | Problemi non risolti sui dati101 |
| 2.2 | Identificazione dei violatori101 |
| 2.3 | Identificazione delle popolazioni di analisi104 |
| 2.4 | Scelta del metodo di replicazione dei valori mancanti 105 |
| 2.5 | Finalizzazione del SAP Vers. 2.0 |
| 2.6 | Consistenza delle codifiche dei termini medici105 |
| 2.7 | Riconciliazione degli Eventi Avversi Seri105 |
| 2.8 | Definizione delle attività propedeutiche al congelamento del DB 105 |
| 2.9 | Decisione di inviare la minuta al CE106 |
| ર | ΔΙΙΕΘΑΤΙ |



Doc code: BIOSTAT.SAP. 02

Pag. 100 of 115

#### 1 INTRODUZIONE

In data 10 Giugno 2020, sulla piattaforma zoom meeting, si è tenuto il "Data Review Meeting" (DRM) dello studio in oggetto. I partecipanti alla riunione sono elencati nella pagina firme. Il DRM si è svolto seguendo le indicazioni delle SOP di Fullcro Srl (CRO incaricata della gestine dello studio) e seguendo le indicazioni del Piano di Analisi Statistica (Statistical Analysis Plan) Versione 1.1 del 4 Giugno 2020.

Gli obiettivi del DRM erano definiti nell'Agenda inviata al Team il 5 Giugno 2020 che si riporta nell'Allegato 1.

Questo documento è strutturato sulla base dei punti elencati nell'Agenda. In particolare, per la definizione delle popolazioni in studio, in Allegato 2 è riportato l'elenco completo. Questa lista sarà inclusa dallo Statistico dello studio in un dataset derivato che farà parte integrante del database clinico.

In ogni sezione del presente documento saranno elencate le decisioni prese dal Team sui vari argomenti. La firma del presente documento certificherà l'accettazione a maggioranza delle decisioni prese.

La minuta del DRM sarà inclusa come allegato del SAP Versione 2.0.

Il giorno 22 Giugno è stata fatta una call, sempre su piattaforma zoom meeting, al fine chiarire alcuni punti emersi durante la revisione della Minuta del DRM. Le decisioni vanno ad integrare il presente documento nella sua versione draft 0.2. Una volta approvato da tutto il team, verrà prodotta la versione finale che sarà inserita nel SAP.



Doc code: BIOSTAT.SAP. 02

Pag. 101 of 115

#### 2 ARGOMENTI IN AGENDA

#### 2.1 Problemi non risolti sui dati

Il primo congelamento del Database è stato fatto in data 5 Giugno 2020. Il System Administrator (SA) della eCRF (electronic Case Report Form) di Fullcro ha revocato tutti I diritti di accesso in scrittura. A seguire è stato fatto un "cleaning" dei dati. Sul Database è emersa una sola inconsistenza:

Tabella: Eventi Avversi

Soggetto: 121

Num. evento: 3

Campo inconsistente: Descrizione

Contunuto: "OARLIC VOICE"

#### **Decisione del Team**

Una volta finalizzata la presente minuta, il PM dello studio richiederà lo scongelamento del Database seguendo le indicazioni della SOP Fullcro dedicata. Il SA rilascerà le credenziali in scrittura al PI per la modifica del dato.

#### 2.2 Identificazione dei violatori

Utilizzando un listato per soggetto, preparato dallo Statistico dello studio, il Team ha esaminato tutte le possibili violazioni al protocollo. Il listato era strutturato per tipologia di violazione:

- 1. Criteri di selezione
- 2. Aderenza
- 3. Uscita prematura dallo studio
- 4. Finestre di accettabilità sulle date visita

Nel corso della riunione sono stati identificati quattro "screening failure", soggetti che, arruolati (visita 0 – screening) non sono stati randomizzati. Questa è la lista:



Doc code: BIOSTAT.SAP. 02

Pag. 102 of 115

Soggetti n.: 055 – 113 – 118 – 195

Questi soggetti sono stati esclusi da tutte le popolazioni di analisi.

Di seguito sono riportati i risultati e le decisioni del Team su ognuna delle quattro categorie.

#### 1 - Criteri di selezione

Non è stata osservata nessuna violazione.

#### **Decisione del Team**

N.A.

#### 2 - Aderenza

Per "aderenza" il Team ha confermato la definizione riportata nel SAP:

considerando il totale dei giorni di studio da V1 a V6 al denominatore e il totale dei giorni di effettivo uso del prodotto oggetto dello studio (derivati dal diario del soggetto) al numeratore per lo stesso nel periodo (es. 45 gg di utilizzo/90 gg da V1 a V6 = 0,50); il soggetto è considerato "aderente" se il risultato è maggiore/uguale a 0,90.

#### **Decisione del Team**

Fissata la soglia del 90%, il Team ha deciso che nel range 70%-90% la violazione del soggetto era MINORE. Sotto la soglia del 70% il soggetto era da considerarsi violatore MAGGIORE.

Nella call del 22 Giugno è stato introdotto un ulteriore criterio per l'identificazione dei violatori. Non sarà considerato violatore MAGGIORE il soggetto che, nonostante abbia aderenza sotto la soglie del 70%, sia un "Continuous Quitter", cioè, non abbia consumeto sigarette convenzionali da Visita 4 a Visita 6. Due soggetti non aderenti sono stati considerati nella popolazione Per-Protocol in quanto da Visita 4 hanno smesso di fumare sigarette convenzionali:



Doc code: BIOSTAT.SAP. 02

Pag. 103 of 115

064; 119

#### Lista delle violazioni MAGGIORI

#### Soggetti numero:

| 004 | 011 | 012 | 015 | 018 | 032 | 036 | 048 | 059 | 066 | 090 | 098 | 115 |
|-----|-----|-----|-----|-----|-----|-----|-----|-----|-----|-----|-----|-----|
| 122 | 124 | 130 | 156 | 162 | 167 | 181 | 188 | 193 | 199 | | | |

#### Lista delle violazioni MINORI

#### Soggetti numero:

002 039 042 080 086 135 136 140 147 149 160 179 212

#### 3 – Uscita prematura dallo studio

Per definizione, tutti i soggetti "drop-out" a Visita 6 sono da ritenersi violatori MAGGIORI. Tutti i soggetti che escono dallo studio dopo Visita 2 sono stati esclusi solo dalla popolazione Per-Protocol. I soggetti che escono dallo studio dopo Visita 1 sono stati esclusi anche dalla popolazione ITT.

Nalla call del 22 Giugno è stato deciso di considerare una seconda popolazione PP, la "Per-Protocol V7", composta da tutti i soggetti, non violatori, che completano anche la visita di follow-up (Visita 7).

#### <u>Decisione del Team</u>

Nessuna osservazione da parte del Team.

<u>Lista delle violazioni MAGGIORI – soggetti non inclusi nella popolazione PP</u>

Soggetti numero:



Doc code: BIOSTAT.SAP. 02

Pag. 104 of 115

012 015 018 048 130 137 163 183 189

<u>Lista delle violazioni MAGGIORI – soggetti non inclusi nella popolazione PPV7</u>

Soggetti numero:

032 090 167 180 034 071 074 077 079 091 095 103 112 115

124 129 184 194 202 206 214

<u>Lista delle violazioni MAGGIORI – soggetti non inclusi nelle popolazioni ITT e PP</u>

Soggetti numero:

015 163 183

#### 4 – Finistre di accettabilità sulle date visita

Il Protocollo prevedeva una finestra di accettabilità sulle date di ogni visita. In dettaglio:

Visita 1: ≤7 giorni rispetto a Visita 0

Visite 2-3-4: ±3 giorni rispetto a Visita 1

Visite 5-6-7: ±7 giorni rispetto a Visita 1

#### <u>Decisione del Team</u>

Dopo un'attenta analisi del listato, considerando la tipologia dello studio, il Team ha ritenuto che le piccole differenze rispetto alle finestre di accettabilità osservate in alcune visite non sono da considerare violazioni.

#### 2.3 Identificazione delle popolazioni di analisi

Utilizzando il listato citato, è stato possibile identificare i soggetti da includere nelle tre popolazioni di analisi. La numerosità delle popolazioni è la seguente:



Doc code: BIOSTAT.SAP. 02

Pag. 105 of 115

Popolazione Safety: 220

Popolazione Intention-To-Treat: 217

Popolazione **Per-Protocol**: 193

Popolazione **Per-Protocol V7**: 177

Il dettaglio per soggetto è riportato in Allegato 2.

#### 2.4 Scelta del metodo di replicazione dei valori mancanti

Per l'analisi inferenziale degli endpoint a risposta, il soggetto drop-out è per definizione un "non Responder" (non quitter/failure). Per gli altri endpoint, come riportato nel Capitolo 5.1 del SAP, il metodo di replicazione dei dati mancanti sarà il LOCF (Last Observation Carried Forward).

#### 2.5 Finalizzazione del SAP Vers. 2.0

Nessuna modifica del SAP Versione 1.1 è stata richiesta per cui la versione 2.0 includerà solamente la sezione "Decisioni prese durante il DRM" e l'allegato "Minuta del DRM" con i suoi allegati.

#### 2.6 Consistenza delle codifiche dei termini medici

Il listato delle codifiche dei termini medici (solo Eventi Avversi) è stato inviato dallo Statistico al Team il 5 Giugno. A parte il termine non codificato (vedi Sezione 2.1) non è stata segnalata nessuna inconsistenza.

#### 2.7 Riconciliazione degli Eventi Avversi Seri

N.A. (nessun Evento Avverso Serio osservato durante lo studio).

#### 2.8 Definizione delle attività propedeutiche al congelamento del DB



Doc code: BIOSTAT.SAP. 02

Pag. 106 of 115

Una volta finalizzata la presente minuta, il PM chiederà lo scongelamento del DB per permettere l'inserimento delle ultime query e la loro risoluzione. Quando il SA avrà verificato la completezza dei dati (data cleaning), si procederà con il secondo congelamento.

#### 2.9 Decisione di inviare la minuta al CE

Al momento il Team ha deciso di non inviare la minuta al CE.

#### 3 ALLEGATI

ALLEGATO 1 Agenda del DRM

ALLEGATO 2 Listato delle popolazioni di analisi



Doc code: BIOSTAT.SAP. 02

Pag. 107 of 115

# **ALLEGATO 1**

# Agenda del DRM



Doc code: BIOSTAT.SAP. 02

Pag. 108 of 115

#### **DATA REVIEW MEETING**

#### 10 June 2020

## (The meeting will be held by conference call)

#### **AGENDA**

- Review of the not already solved problems on the data (pending discrepancies, missing data, other pending issues).
- 2. Identification of the Protocol violations (randomization, Inclusion/Exclusion Criteria, low compliance, other violations).
- **3.** Identification of the analysis populations.
- **4.** Values to replace the missing values (drop-out patients) for the Intention-to-treat analysis.
- **5.** Finalization of the Statistical Analysis Plan (SAP Version 2.0).
- **6.** Consistency check on the coding.
- 7. Review on the possible inconsistencies between the SAEs Data Base and the clinical Data Base still not solved.
- **8.** Definition of all the activities necessary for the Data Base freezing.
- 9. Discussion on the opportunity to send the Data Review Meeting minute and the SAP to the Ethic Committee



Doc code: BIOSTAT.SAP. 02

Pag. 109 of 115

# **ALLEGATO 2**

# Listato delle popolazioni di analisi



Doc code: BIOSTAT.SAP. 02

Pag. 110 of 115

| 01-001<br>01-002 | Υ | Υ | | |
|------------------|---|---|---|---|
| 01-002 | | Ť | Υ | Υ |
| 01-002 | Υ | Υ | Υ | Υ |
| 01-003 | Υ | Υ | Υ | Υ |
| 01-004 | Υ | Υ | N | N |
| 01-005 | Υ | Υ | Υ | Υ |
| 01-006 | Υ | Υ | Υ | Υ |
| 01-007 | Υ | Υ | Υ | Υ |
| 01-008 | Υ | Υ | Υ | Υ |
| 01-009 | Υ | Υ | Υ | Υ |
| 01-010 | Υ | Υ | Υ | Υ |
| 01-011 | Υ | Υ | N | N |
| 01-012 | Υ | Υ | N | N |
| 01-013 | Υ | Υ | Υ | Υ |
| 01-014 | Υ | Υ | Υ | Υ |
| 01-015 | Υ | N | N | N |
| 01-016 | Υ | Υ | Υ | Υ |
| 01-017 | Υ | Υ | Υ | Υ |
| 01-018 | Υ | Υ | N | N |
| 01-019 | Υ | Υ | Υ | Υ |
| 01-020 | Υ | Υ | Υ | Υ |
| 01-021 | Υ | Υ | Υ | Υ |
| 01-022 | Υ | Υ | Υ | Υ |
| 01-023 | Υ | Υ | Υ | Υ |
| 01-024 | Υ | Υ | Υ | Υ |
| 01-025 | Υ | Υ | Υ | Υ |
| 01-026 | Υ | Υ | Υ | Υ |
| 01-027 | Υ | Υ | Υ | Υ |
| 01-028 | Υ | Υ | Υ | Υ |
| 01-029 | Υ | Υ | Υ | Υ |
| 01-030 | Υ | Υ | Υ | Υ |
| 01-031 | Υ | Υ | Υ | Υ |
| 01-032 | Υ | Υ | N | N |
| 01-033 | Υ | Υ | Υ | Υ |
| 01-034 | Υ | Υ | Υ | N |
| 01-035 | Υ | Υ | Υ | Υ |
| 01-036 | Υ | Υ | N | N |
| 01-037 | Υ | Υ | Υ | Υ |
| 01-038 | Υ | Υ | Υ | Υ |
| 01-039 | Υ | Υ | Υ | Υ |
| 01-040 | Υ | Υ | Υ | Υ |



Doc code: BIOSTAT.SAP. 02

Pag. 111 of 115

| 1 1 | | l | 1 | l |
|--------|---|---|---|---|
| 01-041 | Υ | Υ | Υ | Υ |
| 01-042 | Υ | Υ | Υ | Υ |
| 01-043 | Υ | Υ | Υ | Υ |
| 01-044 | Υ | Υ | Υ | Υ |
| 01-045 | Υ | Υ | Υ | Υ |
| 01-046 | Υ | Υ | Υ | Υ |
| 01-047 | Υ | Υ | Υ | Υ |
| 01-048 | Υ | Υ | N | N |
| 01-049 | Υ | Υ | Υ | Υ |
| 01-050 | Υ | Υ | Υ | Υ |
| 01-051 | Υ | Υ | Υ | Υ |
| 01-052 | Υ | Υ | Υ | Υ |
| 01-053 | Υ | Υ | Υ | Υ |
| 01-054 | Υ | Υ | Υ | Υ |
| 01-055 | N | N | N | N |
| 01-056 | Υ | Υ | Υ | Υ |
| 01-057 | Υ | Υ | Υ | Υ |
| 01-058 | Υ | Υ | Υ | Υ |
| 01-059 | Υ | Υ | N | N |
| 01-060 | Υ | Υ | Υ | Υ |
| 01-061 | Υ | Υ | Υ | Υ |
| 01-062 | Υ | Υ | Υ | Υ |
| 01-063 | Υ | Υ | Υ | Υ |
| 01-064 | Υ | Υ | Υ | Υ |
| 01-065 | Υ | Υ | Υ | Υ |
| 01-066 | Υ | Υ | N | N |
| 01-067 | Υ | Υ | Υ | Υ |
| 01-068 | Υ | Υ | Υ | Υ |
| 01-069 | Υ | Υ | Υ | Υ |
| 01-070 | Υ | Υ | Υ | Υ |
| 01-071 | Υ | Υ | Υ | N |
| 01-072 | Υ | Υ | Υ | Υ |
| 01-073 | Υ | Υ | Υ | Υ |
| 01-074 | Υ | Υ | Υ | N |
| 01-075 | Υ | Υ | Υ | Υ |
| 01-076 | Υ | Υ | Υ | Υ |
| 01-077 | Υ | Υ | Υ | N |
| 01-078 | Υ | Υ | Υ | Υ |
| 01-079 | Υ | Υ | Υ | N |
| 01-080 | Υ | Υ | Υ | Υ |
| 01-081 | Υ | Υ | Υ | Υ |
| | | • | | • |



Doc code: BIOSTAT.SAP. 02

Pag. 112 of 115

| 01-082 | Υ | Υ | Υ | Υ |
|--------|---------------|---|---|---|
| 01-083 | Υ | Υ | Υ | Υ |
| 01-084 | Υ | Υ | Υ | Υ |
| 01-085 | Υ | Υ | Υ | Υ |
| 01-086 | Υ | Υ | Υ | Υ |
| 01-087 | Υ | Υ | Υ | Υ |
| 01-088 | Υ | Υ | Υ | Υ |
| 01-089 | Y | Υ | Υ | Υ |
| 01-090 | Y | Υ | N | N |
| 01-091 | <u>.</u><br>Ү | Y | Y | N |
| 01-092 | <u>.</u><br>Ү | Y | Y | Y |
| 01-093 | Υ | Y | Y | Y |
| 01-094 | <u>.</u><br>Ү | Y | Y | Y |
| 01-095 | <u>'</u> | Y | Y | N |
| 01-096 | Y | Y | Y | Y |
| 01-090 | Y | Y | Y | Y |
| 01-097 | Y | Y | N | N |
| 01-098 | Y | Y | Y | Y |
| 01-100 | Y | Y | Y | Y |
| 01-101 | Y | Υ | Y | Y |
| 01-102 | Υ | Y | Y | Y |
| 01-103 | Υ | Y | Y | N |
| 01-104 | Υ | Υ | Υ | Υ |
| 01-105 | Υ | Υ | Υ | Υ |
| 01-106 | Υ | Υ | Υ | Υ |
| 01-107 | Υ | Υ | Υ | Υ |
| 01-108 | Υ | Υ | Υ | Υ |
| 01-109 | Υ | Υ | Υ | Υ |
| 01-110 | Υ | Y | Υ | Υ |
| 01-111 | Υ | Υ | Υ | Υ |
| 01-112 | Υ | Υ | Υ | N |
| 01-113 | N | N | N | Ν |
| 01-114 | Υ | Υ | Υ | Υ |
| 01-115 | Υ | Υ | N | N |
| 01-116 | Υ | Υ | Υ | Υ |
| 01-117 | Υ | Υ | Υ | Υ |
| 01-118 | N | N | N | N |
| 01-119 | Υ | Υ | Υ | Υ |
| 01-120 | Υ | Υ | Υ | Υ |
| 01-121 | Υ | Υ | Υ | Υ |
| 01-122 | Υ | Υ | N | N |



Doc code: BIOSTAT.SAP. 02

Pag. 113 of 115

| 01 122 | V | l v | l v | l v |
|----------|---|-----|-----|-----|
| 01-123 | Y | Y | Y | Y |
| 01-124 | Y | Y | N | N |
| 01-125 | Υ | Y | Y | Y |
| 01-126 | Υ | Y | Υ | Υ |
| 01-127 | Υ | Υ | Υ | Υ |
| 01-128 | Υ | Υ | Υ | Υ |
| 01-129 | Υ | Υ | Υ | N |
| 01-130 | Υ | Υ | N | N |
| 01-131 | Υ | Υ | Υ | Υ |
| 01-132 | Υ | Υ | Υ | Υ |
| 01-133 | Υ | Υ | Υ | Υ |
| 01-134 | Υ | Υ | Υ | Υ |
| 01-135 | Υ | Υ | Υ | Υ |
| 01-136 | Υ | Υ | Υ | Υ |
| 01-137 | Υ | Υ | N | N |
| 01-138 | Υ | Υ | Υ | Υ |
| 01-139 | Υ | Υ | Υ | Υ |
| 01-140 | Υ | Υ | Υ | Υ |
| 01-141 | Υ | Υ | Υ | Υ |
| 01-142 | Υ | Υ | Υ | Υ |
| 01-143 | Υ | Υ | Υ | Υ |
| 01-144 | Υ | Υ | Υ | Υ |
| 01-145 | Υ | Υ | Υ | Υ |
| 01-146 | Υ | Υ | Υ | Υ |
| 01-147 | Υ | Υ | Υ | Υ |
| 01-148 | Υ | Υ | Υ | Υ |
| 01-149 | Υ | Υ | Υ | Υ |
| 01-150 | Υ | Υ | Υ | Υ |
| 01-151 | Υ | Υ | Υ | Υ |
| 01-152 | Υ | Υ | Υ | Υ |
| 01-153 | Υ | Υ | Υ | Υ |
| 01-154 | Υ | Υ | Υ | Υ |
| 01-155 | Υ | Υ | Υ | Υ |
| 01-156 | Υ | Υ | N | N |
| 01-157 | Υ | Υ | Υ | Υ |
| 01-158 | Υ | Υ | Υ | Υ |
| 01-159 | Υ | Υ | Υ | Υ |
| 01-160 | Υ | Υ | Υ | Υ |
| 01-161 | Υ | Υ | Υ | Υ |
| 01-162 | Υ | Υ | N | N |
| 01-163 | Y | N | N | N |
| <u> </u> | • | ., | 1 | |



Doc code: BIOSTAT.SAP. 02

Pag. 114 of 115

| 01-164 | Υ | Υ | Υ | Υ |
|--------|---|---|---|---|
| 01-165 | Υ | Υ | Υ | Υ |
| 01-166 | Υ | Υ | Υ | Υ |
| 01-167 | Υ | Υ | N | N |
| 01-168 | Υ | Υ | Υ | Υ |
| 01-169 | Υ | Υ | Υ | Υ |
| 01-170 | Υ | Υ | Υ | Υ |
| 01-171 | Υ | Υ | Υ | Υ |
| 01-172 | Υ | Υ | Υ | Υ |
| 01-173 | Υ | Υ | Υ | Υ |
| 01-174 | Υ | Υ | Υ | Υ |
| 01-175 | Υ | Υ | Υ | Υ |
| 01-176 | Υ | Υ | Υ | Υ |
| 01-177 | Υ | Υ | Υ | Υ |
| 01-178 | Υ | Υ | Υ | Υ |
| 01-179 | Υ | Υ | Υ | Υ |
| 01-180 | Υ | Υ | Υ | N |
| 01-181 | Υ | Υ | N | N |
| 01-182 | Υ | Υ | Υ | Υ |
| 01-183 | Υ | N | N | N |
| 01-184 | Υ | Υ | Υ | N |
| 01-185 | Υ | Υ | Υ | Υ |
| 01-186 | Υ | Υ | Υ | Υ |
| 01-187 | Υ | Υ | Υ | Υ |
| 01-188 | Υ | Υ | N | N |
| 01-189 | Υ | Υ | N | N |
| 01-190 | Υ | Υ | Υ | Υ |
| 01-191 | Υ | Υ | Υ | Υ |
| 01-192 | Υ | Υ | Υ | Υ |
| 01-193 | Υ | Υ | N | N |
| 01-194 | Υ | Υ | Υ | N |
| 01-195 | N | N | N | N |
| 01-196 | Υ | Υ | Υ | Υ |
| 01-197 | Υ | Υ | Υ | Υ |
| 01-198 | Υ | Υ | Υ | Υ |
| 01-199 | Υ | Υ | N | N |
| 01-200 | Υ | Υ | Υ | Υ |
| 01-201 | Υ | Υ | Υ | Υ |
| 01-202 | Υ | Υ | Υ | N |
| 01-203 | Υ | Υ | Υ | Υ |
| 01-204 | Υ | Υ | Υ | Υ |



Doc code: BIOSTAT.SAP. 02

Pag. 115 of 115

| 01-205 | Υ | Υ | Υ | Υ |
|--------|---|---|---|---|
| 01-206 | Υ | Υ | Υ | N |
| 01-207 | Υ | Υ | Υ | Υ |
| 01-208 | Υ | Υ | Υ | Υ |
| 01-209 | Υ | Υ | Υ | Υ |
| 01-210 | Υ | Υ | Υ | Υ |
| 01-211 | Υ | Υ | Υ | Υ |
| 01-212 | Υ | Υ | Υ | Υ |
| 01-213 | Υ | Υ | Υ | Υ |
| 01-214 | Υ | Υ | Υ | N |
| 01-215 | Υ | Υ | Υ | Υ |
| 01-216 | Υ | Υ | Υ | Υ |
| 01-217 | Υ | Υ | Υ | Υ |
| 01-218 | Υ | Υ | Υ | Υ |
| 01-219 | Υ | Υ | Υ | Υ |
| 01-220 | Υ | Υ | Υ | Υ |
| 01-221 | Υ | Υ | Υ | Υ |
| 01-222 | Υ | Υ | Υ | Υ |
| 01-223 | Υ | Υ | Υ | Υ |
| 01-224 | Υ | Υ | Υ | Υ |